# **Clinical Study Protocol**

A Phase 1, Randomized, Placebo-Controlled, Single Ascending Dose First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VIS649

Administered Intravenously in Healthy Subjects

Sponsor: Visterra Inc.

275 2<sup>nd</sup> Avenue

Waltham, MA 02451

Contract Research Organization: PAREXEL International

Early Phase Clinical Unit-Los Angeles

1560 Chevy Chase Drive, Suite 140

Glendale, CA 91206

**USA** 

Sponsor Study Number: VIS649-101

IMP Name: VIS649

Development Phase: Phase 1 safety and pharmacokinetics

Version (Date) of Final Protocol: Amendment 2, Version 3.0 (Final) (12 Mar 2019)

This clinical study will be conducted in accordance with the International Council for Harmonisation Tripartite Guideline for Good Clinical Practice (GCP) (E6), the protocol and with other applicable regulatory requirements.

#### Confidentiality Statement

This document contains confidential information of Visterra Inc. Do not copy or distribute without written permission from the Sponsor.

#### SIGNATURE PAGE

# Declaration of Sponsor or Responsible Medical Expert

**Protocol Title:** A Phase 1, Randomized, Placebo-Controlled, Single Ascending Dose First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VIS649 Administered Intravenously in Healthy Subjects

This clinical study protocol was subjected to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the investigational medicinal product (IMP), as well as with the moral, ethical and scientific principles governing clinical research as set out in the guidelines on GCP applicable to this clinical study.

## Sponsor Signatory/Responsible Medical Expert



#### SIGNATURE PAGE

#### **Declaration of the Principal Investigator**

**Protocol Title:** A Phase 1, Randomized, Placebo-Controlled, Single Ascending Dose First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VIS649 Administered Intravenously in Healthy Subjects

This clinical study protocol was subjected to critical review and has been released by the Sponsor. The information it contains is consistent with current risk and benefit evaluation of the IMP, as well as with the moral, ethical and scientific principles governing clinical research as set out in the guidelines on GCP applicable to this clinical study.

### Principal Investigator



## LIST OF STUDY STAFF

| Sponsor | Visterra Inc.<br>275 2 <sup>nd</sup> Avenue |
|---|---|
| Principal Investigator | Waltham, MA 02451 Principal Investigator PAREXEL International Early Phase Clinical Unit–Los Angeles 1560 Chevy Chase Drive, Suite 140 Glendale, CA 91206 USA |
| Contract Research Organization | PAREXEL International Early Phase Clinical Unit – Los Angeles 1560 Chevy Chase Drive, Suite 140 Glendale, CA 91206 USA |
| Adverse Event Reporting | PAREXEL Pharmacovigilance Safety Services |
| Medical Monitor | PAREXEL International 2520 Meridian Parkway Durham, NC 27713 USA |
| Clinical Laboratory | GenX Laboratories GenX Laboratories Inc. |
| Bioanalytical Laboratory (PK & ADA) | Syneos Health 301D College Road Princeton, NJ 08540 |

#### PROTOCOL AMENDMENTS

### Protocol Amendment No. 2, dated 12 Mar 2019

The following changes were made to final version 2.0 of the Clinical Study Protocol, dated 20 Dec 2018.

- 1. Cohort 5 was finalized as a cohort (no longer optional), and was amended as such throughout the document.
- 2. The Schedule of Assessments was revised to reflect the specific procedures for cohort 5 including TENIVAC® (tetanus/diphtheria) vaccine administration at Day 28, and necessary serology; a footnote was added to the Schedule of Assessments to indicate these procedures are for cohort 5 only.
- 3. The time points in the Schedule of Assessments were updated to add a Day 31 visit for cohort 5 only.
- 4. A footnote was added to the Schedule of Assessments to indicate that blood sampling for lymphocyte populations and future PD biomarkers is not applicable for cohort 5.
- 5. Background information regarding TENIVAC® was added to the Introduction section and a reference was added.
- 6. Adverse reactions associated with TENIVAC® were added to the Risk-Benefit Assessment.
- 7.
- 8. Study Overview was updated for cohort 5.
- 9. Number of Subjects were revised to describe subjects within cohorts 1-4 and in cohort 5.
- 10. Inclusion and exclusion criteria regarding TENIVAC® were added.
- 11. The Investigational Medicinal Product section was updated to include information regarding toxoid vaccination.
- 12. Randomization numbers were updated as per number of subjects in cohort 5.

- 13. Information for breaking the randomization code was moved to the Randomization Numbers section.
- 14. Measurements and Methods of Assessment was revised to include the most recent vaccination information.
- 15. Clinical Laboratory Assessments was updated to include TENIVAC® serology.
- 16. Total blood volume planned for collection from each subject over the course of the entire study was corrected.
- 17. Under Adverse Event, study drug and vaccine administration sites were specified.
- 18. The Statistical Analysis Plan was specified under Pharmacokinetics/Pharmacodynamics Analyses.
- 19. A separate section in Statistical Methods was included for assessment of response to TENIVAC® vaccination.
- 20. Minor editorial corrections were done throughout.

#### Protocol Amendment No.1, dated 20 Dec 2018.

The following changes were made to final version 1.0 of the Clinical Study Protocol, dated 20 Aug 2018.

- 1. The study design was revised to indicate that back-up subjects who are not randomized into the cohort, but otherwise meet eligibility, may be re-screened after discussion among the Principal Investigator, Medical Monitor, and the Sponsor.
- 2. It was clarified that the Modification of Diet in Renal Disease will be used for the eGFR calculation.
- 3. Timeframe limitations for prescription or over-the-counter medications were clarified.
- 4. Exclusion criteria regarding grapefruit and Seville-oranges were removed.
- 5. A cotinine test at Screening and admission was added.
- 6. It was clarified that the Site 11-panel urine drug screen will also test for methylenedioxymethamphetamine, tricyclic antidepressants, oxycodone, and propoxyphene, and that if a subject tests positive on these 4 tests, inclusion of that subject

into the study will be based on the Principal Investigator's judgment with consultation, if needed, with the Medical Monitor and Sponsor.

- 7. It was revised to indicate that the study drug will be destroyed by carbonization rather than incineration.
- 8. It was revised to indicate that subject weight will be captured after admission to the research unit (Day -1) and will be used by the pharmacy staff for subject-specific dose calculation.
- 9. It was clarified that electrocardiograms will be evaluated by a qualified physician or by a qualified physician's assistant for the presence of abnormalities.
- 10. Individual blood volumes as well as the total amount of blood to be collected over the course of the study were revised.
- 11. The days of collection for pharmacodynamic (lymphocyte populations) were revised (removal of Week 1/Day 7, Week 7/Day 49, and Week 12, Day 84).
- 12. It was clarified that vital signs will be tested at Screening <u>and Day -1</u> and that temperature will be measured at Day -1 and Day 1 (pre-dose only).
- 13. It was clarified that post-dose blood pressure, pharmacodynamics, and safety laboratory data collection should be based on the end of infusion time.
- 14. The term "whole blood" was removed from the phrase "circulating lymphocyte populations."



- 17. Regarding the "changes in circulating lymphocyte populations assessment," it was clarified that this assessment will be done for all lymphocytes, and also for lymphocyte subjects that are noted to show changes from baseline.
- 18. In Section 8.2.3, it was clarified that the PD populations are **safety** subsets.
- 19. AUC<sub>0-112d</sub> and AUC<sub>0-last</sub> were added to the list of PK parameters.

- 20. Where it was appropriate the term "race" was changed to "ethnicity."
- 21. ADA population was removed from the analysis.
- 22. Minor numerical corrections were made to Table 8.
- 23. Minor typographical errors were corrected.

## PROTOCOL SYNOPSIS

| Protocol Title | A Phase 1, Randomized, Placebo-Controlled, Single Ascending Dose First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VIS649 Administered Intravenously in Healthy Subjects |
|---|---|
| Study Numbers | Sponsor Protocol No.: VIS649-101 |
| Development Phase | Phase 1, safety and pharmacokinetics (PK) |
| Sponsor | Visterra Inc. |
| Principal Investigator | |
| Study Center | PAREXEL Early Phase Clinical Unit-Los Angeles |
| Study Objectives | Primary Objective: To evaluate the safety and tolerability of VIS649 in healthy subjects Secondary Objectives: • To characterize the PK profile of VIS649 • To evaluate the effect of ethnicity on the pharmacokinetic (PK) profile of a single intravenously (IV) administered dose of VIS649 in healthy Japanese and non-Japanese subjects • To characterize the levels of anti-drug antibodies • To characterize the effect of VIS649 on pharmacodynamic (PD) parameters including: • changes in serum total IgA, IgG and IgM concentrations and time to recovery • changes in circulating lymphocyte populations in cohorts 1-4 (this assessment will be done for all lymphocytes, and also for lymphocyte subsets that are noted to show changes from baseline). • assess ADA status impact on VIS649 PK parameters |
| Study Design | This is a Phase 1, randomized, placebo-controlled, double-blind, single ascending dose study of IV VIS649 in healthy subjects. Potential subjects will be carefully screened for eligibility prior to study enrollment. Randomization and blinding will occur according to a core randomization list administered by the site's unblinded pharmacist. The study will enroll up to 51 subjects and will be conducted in five |

| | sequential dosing cohorts. Cohorts 1-4 will have four different dose levels (0.5, 2.0, 6.0 and 12 mg/kg respectively), enrolling 9 subjects per cohort. Cohort 5 will be on 6.0 mg/kg only and will enroll up to 15 subjects. Subjects will be randomized to VIS649 or placebo in a ratio of 7:2 (7 active, 2 placebo), except for cohort 5, which will be a ratio of 10:5. Back-up subjects who are not randomized into the cohort, but otherwise meet eligibility, may be re-screened after discussion among the Principal Investigator, Medical Monitor, and the Sponsor. Eligible subjects will report to the Clinical Pharmacology Unit (CPU) at study check-in (Day -1) and will be required to stay in the CPU until Day 2 (24 hours post infusion). On Day 1, a single dose of VIS649 or placebo will be administered IV in the morning after a light meal (as per the clinical unit standard). Pharmacokinetics sampling will occur on Day 1 starting with a collection prior to the start of infusion, at the end of infusion (60 minutes), and at 2 hours, 8 hours and 24 hours post end of infusion. All subjects will have PK samples drawn on Days 1-3, 7, 14, 28, 42, 56, 70, and 112. Pharmacodynamics sampling (serum immunoglobulin levels) will occur at baseline, Day 3 and weekly thereafter through the Week 8 visit, then once every two weeks through Week 16 (i.e., Weeks 10, 12, 14, and 16). Sentinel subjects will be utilized in cohorts 1-4; the first two subjects in each cohort will be randomized to receive either VIS649 (n=1) or placebo (n=1) and will receive study drug at least 24 hours before the remaining subjects in the cohort (7 subjects) are dosed. These 2 subjects shall remain confined to the study center for 24 hours after study drug administration. The safety profile of these subjects over the 24-hour post-administration period will be reviewed to determine whether it is appropriate to proceed with enrollment of the remaining subjects in the cohort as planned. This will occur for each dose escalation. The remaining 7 subjects in cohorts 1-4 wil |
|---|---|
| | for individual subjects will be approximately 20 weeks (5 months) with the possibility to extend up to 28 weeks (7 months). Each subject will participate in a Screening period lasting 1 to 28 days (0 to 4 weeks), an in-house stay for 2 to 3 days, and a post-administration period of 16 weeks. The scheduled final visit will occur 16 weeks post-dosing (112 days); however, two additional follow-up visits may be performed, at Weeks 20 and 24 post-dosing, if serum immunoglobulins have not returned to>lower limits of normal by the Week 16 visit or if emerging trial data suggest a value of later follow-up (i.e., for detection of anti-drug antibody responses). |
| Investigational Medicinal Product (IMP) | A single dose of VIS649 administered IV over approximately one hour, at four different dose levels: 0.5, 2.0, 6.0 and 12 mg/kg respectively, with a fifth cohort, to receive a 6.0 mg/kg single dose of VIS649 administered intravenously on Day 1 in one arm and a single intramuscular injection of TENIVAC® vaccine on Day 28 into the opposite arm. |
| Number of Subjects | Up to 51 subjects may be enrolled. A total of 16 Japanese subjects (4 subjects each in cohorts 1-4) and 20 non-Japanese subjects (up to 5 subjects each in cohorts 1-4) may be enrolled and randomized to receive a single dose of VIS649 or placebo. No more than one Japanese subject per cohort may be randomized to receive placebo in cohorts 1-4. Up to 15 subjects are expected to be enrolled in cohort 5 with targeted but non-mandatory enrollment of up to 5 Japanese subjects. No more than two Japanese subjects may be randomized to receive placebo in cohort 5. |

| Criteria for Evaluation Safety Endpoints The proportion of subjects with adverse events (AEs) and serious advevents (SAEs) following administration of VIS649; safety will be asses from the time of study drug administration to the end-of-study participati The following safety variables will be assessed from the time of study administration to the end-of-study participation: Adverse event assessments Clinical laboratory tests (hematology, clinical chemistry and urinalyse) Vital signs (sitting blood pressure, pulse, body temperature respiratory rate) 12-lead electrocardiogram (ECG) Adjunctive procedures Physical examination Secondary Endpoints Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as approprive Cmax: Maximum serum VIS649 concentration determined directly the concentration-time profile Tmax: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112 AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration t <sub>1/2</sub> : Apparent terminal elimination half-life Vd: Apparent volume of distribution CL: Apparent volume of distribution |
|---|
| events (SAEs) following administration of VIS649; safety will be assess from the time of study drug administration to the end-of-study participation: The following safety variables will be assessed from the time of study administration to the end-of-study participation: Adverse event assessments Clinical laboratory tests (hematology, clinical chemistry and urinaly: Vital signs (sitting blood pressure, pulse, body temperature respiratory rate) 12-lead electrocardiogram (ECG) Adjunctive procedures Physical examination Secondary Endpoints Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as approprive Cmax: Maximum serum VIS649 concentration determined directly the concentration-time profile Tmax: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile AUC <sub>0-inf</sub> : Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time AUC 0-last: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration t <sub>1/2</sub> : Apparent terminal elimination half-life Vd: Apparent volume of distribution |
| administration to the end-of-study participation: Adverse event assessments Clinical laboratory tests (hematology, clinical chemistry and urinally. Vital signs (sitting blood pressure, pulse, body temperature respiratory rate) 12-lead electrocardiogram (ECG) Adjunctive procedures Physical examination Secondary Endpoints Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as appropriate to concentration-time profile T <sub>max</sub> : Time of maximum serum VIS649 concentration determined directly from the concentration-time profile AUC <sub>0-inf</sub> : Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time AUC <sub>0-last</sub> : Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112 AUC <sub>0-last</sub> : Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration t <sub>1/2</sub> : Apparent terminal elimination half-life Vd: Apparent volume of distribution |
| <ul> <li>Clinical laboratory tests (hematology, clinical chemistry and urinally.</li> <li>Vital signs (sitting blood pressure, pulse, body temperature respiratory rate)</li> <li>12-lead electrocardiogram (ECG)</li> <li>Adjunctive procedures</li> <li>Physical examination</li> <li>Secondary Endpoints</li> <li>Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints</li> <li>The following PK parameters for VIS649 will be determined, as approprioused to Communicate the concentration-time profile</li> <li>Times: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile</li> <li>AUCO-inf: Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time</li> <li>AUC 0-1124: Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112</li> <li>AUC 0-last: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| <ul> <li>Vital signs (sitting blood pressure, pulse, body temperature respiratory rate)</li> <li>12-lead electrocardiogram (ECG)</li> <li>Adjunctive procedures</li> <li>Physical examination</li> <li>Secondary Endpoints</li> <li>Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as appropring the concentration-time profile</li> <li>T<sub>max</sub>: Maximum serum VIS649 concentration determined directly the concentration-time profile</li> <li>T<sub>max</sub>: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile</li> <li>AUC<sub>0-inf</sub>: Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time</li> <li>AUC <sub>0-112d</sub>: Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112</li> <li>AUC <sub>0-last</sub>: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| respiratory rate) • 12-lead electrocardiogram (ECG) • Adjunctive procedures • Physical examination Secondary Endpoints • Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as appropring the concentration-time profile • T <sub>max</sub> : Maximum serum VIS649 concentration determined directly the concentration-time profile • T <sub>max</sub> : Time of maximum serum VIS649 concentration determined directly from the concentration-time profile • AUC <sub>0-inf</sub> : Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time • AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112 • AUC <sub>0-last</sub> : Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration • t <sub>1/2</sub> : Apparent terminal elimination half-life • Vd: Apparent volume of distribution |
| <ul> <li>Adjunctive procedures</li> <li>Physical examination</li> <li>Secondary Endpoints</li> <li>Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as approprious Cmax: Maximum serum VIS649 concentration determined directly the concentration-time profile</li> <li>Tmax: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile</li> <li>AUC0-inf: Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time</li> <li>AUC 0-112d: Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112</li> <li>AUC 0-last: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| <ul> <li>Physical examination Secondary Endpoints <ul> <li>Characterization of anti-drug antibodies (ADA) levels</li></ul></li></ul> |
| <ul> <li>Secondary Endpoints</li> <li>Characterization of anti-drug antibodies (ADA) levels Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as appropriate the concentration-time profile</li> <li>T<sub>max</sub>: Maximum serum VIS649 concentration determined directly the concentration-time profile</li> <li>T<sub>max</sub>: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile</li> <li>AUC<sub>0-inf</sub>: Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time</li> <li>AUC <sub>0-112d</sub>: Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112</li> <li>AUC <sub>0-last</sub>: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| <ul> <li>Characterization of anti-drug antibodies (ADA) levels <i>Pharmacokinetics Endpoints</i> The following PK parameters for VIS649 will be determined, as appropried to Cmax: Maximum serum VIS649 concentration determined directly the concentration-time profile <ul> <li>Tmax: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile</li> <li>AUC<sub>0-inf</sub>: Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time</li> </ul> </li> <li>AUC <sub>0-112d</sub>: Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112</li> <li>AUC <sub>0-last</sub>: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| Pharmacokinetics Endpoints The following PK parameters for VIS649 will be determined, as appropriate the concentration-time profile • T <sub>max</sub> : Maximum serum VIS649 concentration determined directly the concentration-time profile • T <sub>max</sub> : Time of maximum serum VIS649 concentration determined directly from the concentration-time profile • AUC <sub>0-inf</sub> : Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time • AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112 • AUC <sub>0-last</sub> : Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration • t <sub>1/2</sub> : Apparent terminal elimination half-life • Vd: Apparent volume of distribution |
| The following PK parameters for VIS649 will be determined, as appropriate the concentration-time profile • T <sub>max</sub> : Maximum serum VIS649 concentration determined directly the concentration-time profile • T <sub>max</sub> : Time of maximum serum VIS649 concentration determined directly from the concentration-time profile • AUC <sub>0-inf</sub> : Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time • AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112 • AUC <sub>0-last</sub> : Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration • t <sub>1/2</sub> : Apparent terminal elimination half-life • Vd: Apparent volume of distribution |
| <ul> <li>C<sub>max</sub>: Maximum serum VIS649 concentration determined directly the concentration-time profile</li> <li>T<sub>max</sub>: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile</li> <li>AUC<sub>0-inf</sub>: Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time</li> <li>AUC<sub>0-112d</sub>: Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112</li> <li>AUC<sub>0-last</sub>: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| the concentration-time profile T <sub>max</sub> : Time of maximum serum VIS649 concentration determ directly from the concentration-time profile AUC <sub>0-inf</sub> : Area under the concentration-time curve from pre-dose (0) extrapolated to infinite time AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112 AUC <sub>0-last</sub> : Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration t <sub>1/2</sub> : Apparent terminal elimination half-life Vd: Apparent volume of distribution |
| directly from the concentration-time profile • AUC <sub>0-inf</sub> : Area under the concentration-time curve from pre-dose ( 0) extrapolated to infinite time • AUC <sub>0-112d</sub> : Area under the concentration-time curve from pre-dose ( 0) to the concentration on Day 112 • AUC <sub>0-last</sub> : Area under the concentration-time curve from pre-dose ( 0) to the last quantifiable concentration • t <sub>1/2</sub> : Apparent terminal elimination half-life • Vd: Apparent volume of distribution |
| <ul> <li>• AUC <sub>0-112d</sub>: Area under the concentration-time curve from pre-dose (0) to the concentration on Day 112</li> <li>• AUC <sub>0-last</sub>: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>• t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>• Vd: Apparent volume of distribution</li> </ul> |
| <ul> <li>0) to the concentration on Day 112</li> <li>AUC <sub>0-last</sub>: Area under the concentration-time curve from pre-dose (0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| <ul> <li>0) to the last quantifiable concentration</li> <li>t<sub>1/2</sub>: Apparent terminal elimination half-life</li> <li>Vd: Apparent volume of distribution</li> </ul> |
| Vd: Apparent volume of distribution |
| • CI: Apparent clearance |
| CL. Apparent clearance |
| Pharmacodynamics Endpoints |
| • Changes in total serum IgG, IgA and IgM concentrations and time recovery |
| • Changes in circulating lymphocyte populations in cohorts 1-4 only assessment will be done for all lymphocytes, and also for lymphocyte sul |
| that are noted to show changes from baseline). |
| Statistical Methods Sample Size Considerations |
| As this is a first-in-human (FIH) study and no clinical data are available |

formal sample size calculations have been performed. A total of up to 51 evaluable subjects is considered suitable to achieve the study objectives.

Data Presentation/Descriptive Statistics

In general, descriptive statistics for continuous variables will be summarized by treatment group using number of subjects, arithmetic mean, standard deviation, median, minimum and maximum; descriptive statistics for categorical data will be summarized by treatment group using frequency counts and percentages.

Summary of demographics and safety data will be analyzed using descriptive statistics as appropriate.

The VIS649 serum concentrations will be listed and summarized by dose and time point. Individual and mean VIS649 concentration-time profiles will be plotted in linear and semi-log scales. Non-compartmental PK data analysis will be performed for VIS649 treated subjects to estimate the AUC 0-112d, AUC 0-last, AUC0-inf, Cmax, Tmax, t½, CL and Vd. Descriptive statistics for PK parameters will include number of observations, arithmetic mean, standard deviation, arithmetic coefficient of variation (%CV), and geometric mean, median, geometric %CV, minimum and maximum.

The number and percentage of subjects that are ADA positive will be summarized by dose. The impact of ADA on PK and the association with treatment-emergent adverse events and treatment-emergent serious adverse events will be assessed.

PD data will be assessed using change from baseline data and % change from baseline, as appropriate. The PK/PD relationship between investigational medicinal product exposure and exploratory endpoints may also be analyzed by graphical displays if Sponsor requests. Data from cohorts 1-4 will be analyzed separately from cohort 5.

All demographic, safety, PK, and PD data will be listed. Full details of the data analysis will be provided in a separate statistical analysis plan.

## TABLE OF CONTENTS

|-----------------------------------------------|----|
| LIST OF STUDY STAFF | 4 |
| PROTOCOL SYNOPSIS | 5 |
| TABLE OF CONTENTS | 8 |
| LIST OF STUDY STAFF | 4 |
| PROTOCOL AMENDMENTS | 5 |
| PROTOCOL SYNOPSIS | 9 |
| TABLE OF CONTENTS | |
| List of Tables. | 17 |
| List of Figures | 17 |
| LIST OF ABBREVIATIONS AND DEFINITION OF TERMS | 18 |
| 1. INTRODUCTION | 21 |
| 1.1. Background | 21 |
| 1.2. Rationale for the Clinical Study | 24 |
| 1.3. Risk-benefit Assessment | 24 |
| 2. STUDY OBJECTIVES | 28 |
| 2.1. Primary Objective | 28 |
| 2.2. Secondary Objectives | 28 |
| 2.3. Exploratory Objectives | 28 |
| 3. OVERALL DESIGN AND PLAN OF THE STUDY | 29 |
| 3.1. Overview | 29 |
| 3.2. Endpoints | 33 |
| 3.2.1. Primary Endpoint | 33 |

| 3.2 | 2.2. Sec | condary Endpoints | 33 |
|---|---|---|---|
| : | 3.2.2.1. | Pharmacokinetics Endpoints. | 33 |
| | 3.2.2.2. | Pharmacodynamics Endpoints | 34 |
| | 3.2.2.3. | Exploratory Endpoints | 34 |
| 3.3. | Justifica | ation of the Study Design | 34 |
| 3.4. | Stoppin | g Criteria for the Clinical Study and Dose Escalation Criteria | 35 |
| 4. ST | TUDY PO | PULATION | 37 |
| 4.1. | Number | of Subjects | 37 |
| 4.2. | Inclusio | n Criteria | 37 |
| 4.3. | Exclusi | on Criteria | 39 |
| 4.4. | Subject | Withdrawal and Replacement | 41 |
| 4.5. | Termina | ation of the Clinical Study | 42 |
| 5. IN | VESTIGA | ATIONAL MEDICINAL PRODUCT AND TOXOID VACCINATION | 43 |
| 5.1. | Identity | of the Investigational Medicinal Products | 43 |
| 5.2. | Tetanus | /Diphtheria Toxoid Vaccine (TENIVAC®) | 43 |
| 5.3. | Rationa | le for Starting Dose and Dose Escalation | 43 |
| 5.4. | Supply, | Packaging, Labeling and Storage | 46 |
| 5.5. | Drug A | ccountability, Dispensing and Destruction | 46 |
| 5.6. | Subject | Identification and Randomization | 47 |
| 5.6 | 5.1. Sci | eening Numbers | 47 |
| 5.6 | 6.2. Ra | ndomization Numbers | 47 |
| 5.7. | Admini | stration of Investigational Medicinal Products | 48 |
| 5.8. | Compli | ance | 48 |
| 5.9. | Blindin | g and Breaking the Blind | 48 |
| 5.10. | . Prior | and Concomitant Medications | 49 |
| 5.11. | . Treat | ment of Overdose | 49 |
| 6. M | EASURE | MENTS AND METHODS OF ASSESSMENT | 50 |
| 6.1. | Medica | History, Demographic and Other Baseline Information | 50 |

| 6.2. Safety | Variables | 51 |
|-------------|-------------------------------------|----|
| 6.2.1. A | Adverse Events | 51 |
| 6.2.1.1. | Definitions | 51 |
| 6.2.1.2. | Recording of Adverse Events | 53 |
| 6.2.1.3. | Assessment of Adverse Events | 53 |
| 6.2.1.4. | Reporting of Serious Adverse Events | 54 |
| 6.2.1.5. | Follow-up of Adverse Events | 56 |
| 6.2.1.6. | Pregnancy | 56 |
| 6.2.2. C | Clinical Laboratory Assessments | 57 |
| 6.2.2.1. | Anti-drug Antibody Response | 59 |
| 6.2.3. V | Vital Signs | 59 |
| 6.2.4. S | tandard 12-lead Electrocardiograms | 60 |
| 6.2.5. P | hysical Examinations | 60 |
| 6.3. Pharm | nacokinetics Variables | 60 |
| 6.3.1. B | Blood Sample Collection | 60 |
| 6.4. Pharm | nacodynamics Variables | 61 |
| 6.5. Total | Amount of Blood | 61 |
| 7. STUDY C | ONDUCT | 63 |
| 7.1. Sched | lule of Assessments | 63 |
| 7.2. Order | of Assessments | 68 |
| 7.3. Early | Termination | 68 |
| 7.4. End-o | f-Study | 68 |
| 7.5. Restri | ctions | 68 |
| 7.5.1. D | Dietary and Fluid Restrictions | 68 |
| 7.5.2. C | Other Restrictions | 69 |
| 8. STATIST | ICAL METHODS | 70 |
| 8.1. Determ | mination of Sample Size | 70 |
| 8.2. Study | Population | 70 |

| | 8.2. | 1. Disposition of Subjects | 70 |
|---|---|---|---|
| | 8.2. | 2. Protocol Deviations | 70 |
| | 8.2. | 3. Analysis Populations | 70 |
| | 8.3. | General Considerations | 71 |
| | 8.4. | Demographic and Anthropometric Information and Baseline Characteristics | 71 |
| | 8.5. | Prior and Concomitant Medication | 71 |
| | 8.6. | Drug Administration | 72 |
| | 8.7. | Safety Analyses | 72 |
| | 8.7. | 1. Adverse Events | 72 |
| | 8.7. | 2. Clinical Laboratory Tests | 72 |
| | 8.7. | 3. Vital Signs | 72 |
| | 8.7. | 4. Standard 12-lead Electrocardiogram | 73 |
| | 8.7. | 5. Physical Examination | 73 |
| | 8.8. | Pharmacokinetics Analyses | 73 |
| | 8.9. | Pharmacodynamics Analyses | 73 |
| | 8.10. | Pharmacokinetics/Pharmacodynamics Analyses | 74 |
| | 8.11. | Immunogenicity Data (Antibody to VIS649) | 74 |
| | 8.12. | Assessment of Response to Tetanus and Diphtheria Vaccination | 74 |
| | 8.13. | Interim Data Reviews | 74 |
| 9 | ETI | HICAL, LEGAL AND ADMINISTRATIVE ASPECTS | 76 |
| | 9.1. | Data Quality Assurance | 76 |
| | 9.2. | Institutional Review Board | 76 |
| | 9.3. | Access to Source Data/Documents | 76 |
| | 9.4. | Archiving Study Documents | 77 |
| | 9.5. | Good Clinical Practice | 77 |
| | 9.6. | Informed Consent | 78 |
| | 9.7. | Protocol Approval and Amendment(s) | 78 |
| | 9.8. | Confidentiality Data Protection | 79 |

| 9.9. | Publication Policy | 79 |
|---|---|---|
| 10. RF | EFERENCE LIST | 80 |
| List of Ta | ables | |
| Table 1 | Serum Immunoglobulin Normal Ranges, Inclusion Criteria, Predicted M | aximal |
| Nadirs, aı | nd Stopping Rule Thresholds | 27 |
| Table 2 | Cohorts and Dose Administration | 31 |
| Table 3 | Identity of Investigational Products | 43 |
| Table 4 | Identity of Toxoid Vaccination. | 43 |
| Table 5 | Safety margins for targeted clinical doses | 46 |
| Table 6 | Randomization Numbers and Treatment Assignment | 47 |
| Table 7 | Assessment of Relationship of Adverse Events to Investigational Product | 54 |
| Table 8 | Clinical Laboratory Assessments | 58 |
| Table 9 | Approximate Total Amount of Blood for Each Subject | 62 |
| Table 10 | Schedule of Assessments | 64 |
| List of Fi | igures | |
| Figure 1 | Study Flow Chart – Single Ascending Dose Design | 32 |
| Figure 2 | Rationale for VIS649 Starting Dose | 45 |

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation | Definition |
|---|---|
| ADA | Anti-drug antibody |
| AE | Adverse event |
| a-g IgA | Aberrantly glycosylated IgA (synonymous with GD IgA) |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| APRIL | A Proliferation Inducing Ligand |
| AST | Aspartate aminotransferase |
| AUC <sub>0-inf</sub> | Area under the concentration-time curve from pre-dose (time |
| | 0) extrapolated to infinite time $(AUC_{last} + C_{last}/\lambda_z)$ |
| AUC <sub>0-112d</sub> | Area under the concentration-time curve from pre-dose |
| | (time 0) to the concentration on Day 112 |
| AUC <sub>0-last</sub> | Area under the concentration-time curve from pre-dose |
| | (time 0) to the last quantifiable concentration |
| BMI | Body mass index |
| BP | Blood pressure |
| bpm | Beats per minute |
| BUN | Blood Urea Nitrogen |
| CL | Apparent clearance |
| C <sub>max</sub> | Maximum serum concentration |
| CPU | Clinical Pharmacology Unit |
| CRO | Clinical Research Organization |
| CSR | Clinical Study Report |
| CV | Coefficient of variation |
| CVID | Common variable immunodeficiency |
| DBP | Diastolic blood pressure |
| ECG | Electrocardiogram |
| FDA | United States Food and Drug Administration |
| Fe | Percentage of drug excreted unchanged in the urine |
| FIH | First-in-human |
| FSH | Follicle stimulating hormone |
| GCP | Good Clinical Practice |

| GD IgA | Galactose deficient IgA (synonymous with a-g IgA) |
|--------|---------------------------------------------------------|
| GLP | Good Laboratory Practice |
| GMR | Geometric Mean Ratio |
| hCG | Human Chorionic Gonadotropin |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human Immunodeficiency Virus |
| HBsAg | Hepatitis B surface antigen |
| IB | Investigator's Brochure |
| ICD | Informed consent document |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| Ig | Immunoglobulin |
| IgA | Immunoglobulin A |
| IgAN | IgA nephropathy |
| IgG | Immunoglobulin G |
| IgM | Immunoglobulin M |
| IMP | Investigational medicinal product |
| IND | Investigational New Drug |
| IRB | Institutional Review Board |
| KLH | Keyhole limpet hemocyanin |
| mAb | Monoclonal Antibody |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MID | Minimum Intolerable Dose |
| MTD | Maximum tolerated dose |
| NOAEL | No-observed-adverse-effect level |
| OTC | Over-the-counter |
| PD | Pharmacodynamics |
| PK | Pharmacokinetics |
| PT | Preferred Term |
| QTcF | QT interval corrected for heart rate using Fridericia's |
| | correction |
| RR | Respiratory rate |
| SAE | Serious adverse event |
| SBP | Systolic blood pressure |

| SID | Subject identification |
|---|---|
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| SOP | Standard operating procedure |
| TACI | Transmembrane activator and CAML interactor |
| Td | Tetanus/diphtheria |
| TENIVAC® | Trade name for a commercially available tetanus/diphtheria |
| | toxoid vaccine |
| t½ | Terminal elimination half-life |
| T <sub>max</sub> | Time of maximum serum concentration |
| US | United States |
| ULN | Upper level of normal |
| Vd | Apparent volume of distribution |
| WBC | White Blood Cells |
| WHO | World Health Organization |

#### 1. INTRODUCTION

### 1.1. Background

VIS649 is a humanized immunoglobulin G (IgG<sub>2</sub>) monoclonal antibody that binds to and blocks the biological actions of the B-cell growth factor, APRIL (<u>A Proliferation Inducing Ligand</u>), preventing binding to its receptors, transmembrane activator and CAML interactor (TACI) and B-cell maturation antigen (BCMA). Through these receptor interactions, APRIL regulates B-cell mediated immune responses through several mechanisms, including the induction of class switch recombination as well as promotion of plasma cell survival.



VIS649 binds human APRIL with picomolar affinity/avidity as measured by antigen-binding enzyme-linked immunosorbent assay using recombinant trimeric APRIL. VIS649 blocks recombinant APRIL-APRIL receptor interactions, thereby inhibiting APRIL-mediated signaling and B-cell proliferation. VIS649 also binds cynomolgus monkey APRIL, with similar affinity and inhibition of APRIL mediated signaling in both species. The physiological and toxicological effects of VIS649 were therefore evaluated in cynomolgus monkeys, in three preclinical studies.

In an initial non- Good Laboratory Practice (non-GLP) *in-vivo* toxicology study, weekly administration of IV VIS649 at a dose of 25 mg/kg for 8 weeks resulted in an approximately 70% reduction in serum IgA levels (in comparison with control animals) with minimal effect on serum IgM, and an approximately 40% reduction in serum IgG levels. Hematology assessment did not reveal significant perturbation in white blood cell (WBC), lymphocyte, or leukocyte counts and there were no significant differences between treatment groups noted in the peripheral blood and tissue immune profiling, which included markers for total T cells, helper T



These studies led to the conduct of a United States Food and Drug Administration (US FDA) GLP-compliant 4-week repeat-dose IV toxicology study of VIS649 in cynomolgus monkeys, with a 20-week recovery period. Monkeys received weekly VIS649 injections for 4 weeks, at doses of 0 mg/kg (control), 25 mg/kg, 50 mg/kg, or 100 mg/kg.

VIS649-related reductions in total serum IgA levels were observed in all VIS649-treated animals and the reductions were reversible as trends towards return to baseline were observed at all doses. All 3 dose levels demonstrated maximal pharmacologic effect that were consistent with previous studies in reduction in serum IgA and IgG levels with a minimal effect on IgM levels in VIS649 treated animals in comparison to the controls.

Serum IgG levels were moderately reduced,
, for a majority of animals at all timepoints. Serum IgM concentrations did not differ significantly between groups, including control animals.

There was no effect of VIS649 on measured plasma cytokine concentrations in the monkey toxicology studies (nor did VIS649 stimulate significant cytokine release in an *in vitro* human peripheral blood lymphocyte cytokine release assay).

To test the effect of VIS649 on de-novo humoral immune responses to a novel (T-cell dependent) antigen challenge, monkeys were vaccinated with keyhole limpet hemocyanin (KLH)

at Day 7 during dosing, with measurement of KLH-specific IgG and IgM levels through 21 days post immunization. The kinetics of IgM and IgG responses were similar between VIS649 treated and control animals, with moderate suppression of KLH-specific IgG levels which was consistent with the non-specific suppression seen in total IgG levels.



The relatively selective and reversible effect of VIS649 on serum immunoglobulin levels with maximal (but not completely suppressive) effect on IgA suggests that APRIL inhibition may be uniquely suited as a therapeutic strategy for IgA nephropathy.

Further details can be found in the IB [2].

TENIVAC® is a vaccine indicated for active immunization for the prevention of tetanus and diphtheria in persons 7 years of age and older. Vaccines such as TENIVAC® that are comprised of tetanus and diphtheria toxoids are referred to as Td vaccines. Tetanus and diphtheria vaccination is recommended for all adults, with the Centers for Disease Control and Prevention (CDC) Advisory Committee on Immunization Practices advising that individuals without contraindication receive booster tetanus immunization (with tetanus toxoid or tetanus/diphtheria combined toxoid vaccination every ten years. Additional details can be found in the 2018 Recommended Immunization Schedule for Adults Aged 19 Years or Older, United States, 2018. Further details regarding TENIVAC®, specifically, can be found in the full prescribing information. [11].

In this study, TENIVAC® will be used as a vaccine challenge to evaluate the effect of VIS649 on recipients' ability to generate an effective response to antigen exposure, as measured by anti-tetanus toxoid and anti-diphtheria toxoid IgG and IgM responses.

#### 1.2. Rationale for the Clinical Study

This FIH study will assess the safety and tolerability, pharmacokinetics (PK)/pharmacodynamics (PD) of VIS649, a humanized IgG<sub>2</sub> mAb that binds to and blocks the biological actions of the B-cell growth factor, APRIL.

The study is being conducted to establish a dose range that is well tolerated by the majority of study subjects and to provide exploratory data on the potential for the treatment of IgAN, an autoimmune glomerulonephritis characterized by the deposition of IgA-containing immune complexes in the kidney. The results of the clinical study will inform the design and dose selection of subsequent studies.

#### 1.3. Risk-benefit Assessment

While VIS649 has not been evaluated in humans, the known effects of mAbs in humans suggest the following potential toxicities for single dose administration:

- 1. Infusion reactions: Anaphylaxis, fever, chills, rigors, nausea, vomiting, pain, headache, dizziness, shortness of breath, bronchospasm, hypotension, hypertension, pruritus, rash, urticaria, angioedema, diarrhea, tachycardia, and chest pain
- 2. Delayed allergic reactions: Serum sickness (i.e., urticaria, fever, general glandular enlargement, joint pains)
- 3. General: Injection site reaction

Mechanism based potential toxicities that might be anticipated based on VIS649 mechanism of action and preclinical studies include:

**IgA suppression risks**: VIS649 treatment is expected to reduce human IgA levels, with a predicted maximal reduction (with repeated dosing) to approximately 75% below baseline. In this single-ascending dose study, this degree of suppression is unlikely to be achieved, but it is anticipated that at least in the higher dose cohorts, IgA levels will be reduced below baseline, with effect persisting over weeks.

The normal range for serum IgA is approximately 70 to 400 mg/dL in adults

Selective IgA deficiency (defined as persistently undetectable IgA, the most common inherited immunodeficiency syndrome (occurring in about 1 in 500 Caucasian individuals). []. While this condition has heretofore been considered generally benign and is asymptomatic in the majority of patients, there is increasing recognition that selective IgA deficiency may be associated with recurrent sinopulmonary infection, allergy, autoimmunity and gastrointestinal microbiome perturbation [4, 5]. The risk for occurrence of these complications in the current study is low for multiple reasons: 1) IgA is expected to be suppressed, but not reduced to undetectable levels, 2) in this single dose-study, the effects on IgA levels are expected to be transient, and 3) the syndrome of selective IgA deficiency is often associated with additional immunologic impairments including T-cell disorders and common variable immunodeficiency syndrome.

**IgG suppression risks:** VIS649 is expected to have a moderate effect on serum IgG levels (with approximately 40% suppression-below-baseline nadir values predicted).

The normal range for serum IgG is approximately 600 to 1600 mg/dL in adults,

immunodeficiency common variable (CVID), also known acquired as hypogammaglobulinemia, total IgG levels are typically below 250 mg/dL with median values at diagnosis in two recent US cohort studies of 210 mg/dL and 120 mg/dL, respectively [6]. The condition is of heterogenous origin, with loss of function mutations in an APRIL receptor, TACI, identified as one causal association [7]. Proposed diagnostic criteria for CVID include: presence of hypogammaglobulinemia plus a history of recurrent or chronic infection or autoimmunity and with associated IgA deficiency or IgM [8]. Common variable immunodeficiency is associated with recurrent deficiency otitis media, chronic sinusitis, and recurrent pneumonia often resulting in bronchiectasis [9]. Longitudinal studies have demonstrated high rates of lymphoma and diseases of autoimmunity [10]. The risk of these complications in the current study is considered quite low, given the moderate and transient reductions in IgG levels that are anticipated.

**Non-specific immunosuppression risks:** In preclinical toxicology studies, de-novo humoral immune responses to a novel antigen were not suppressed, and peripheral blood myeloid cell line

populations were unaffected. However, there is the possibility of non-specific immunodeficiency with potential risk of exacerbation of pre-existing latent infection or poor response to new infection. These risks are considered minimal due to the single-dose design of this trial, and the expected transient nature of effects.

Pharmacodynamic data including measurement of changes in serum IgG, IgA, and IgM levels in relation to VIS649 exposure will provide valuable information for refinement of the human PK/PD model and selection of appropriate doses for a repeat-dose study. Predicted maximal effects on serum IgG, IgA and IgM levels versus normal range, inclusion criteria thresholds, and stopping rule IG thresholds are summarized in Table 1.

Table 1 Serum Immunoglobulin Normal Ranges, Inclusion Criteria, Predicted Maximal Nadirs, and Stopping Rule Thresholds

| Immunoglobulin<br>Class | Serum<br>Concentration<br>Normal Range<br>in Adults <sup>1</sup> |
|---|---|
| IgA | 66-433 mg/dL<br>[0.66-4.33 g/L] |
| IgG | 635-1741 mg/dL<br>[6.35-17.41 g/L] |
| IgM | 45-281 mg/dL<br>[0.45-2.81 g/L] |

<sup>&</sup>lt;sup>1</sup> Immunoglobulin reference ranges for healthy adult volunteers from the laboratory performing these tests for the study (GenX Lab), as measured with a Beckman Coulter Analyzer, instrument AU480.



There will be no direct health benefit for healthy subjects from receipt of the study drug. The protocol has been designed to minimize the risk to research participants. Subjects will be monitored to detect adverse events (AE)s during the study and followed appropriately to ensure resolution of AEs. Sentinel dosing will be employed within each cohort, and available blinded safety data will be assessed after each dose level to determine if it is safe to escalate to the next planned dose.

TENIVAC® has been associated with the following adverse reactions:

- The most frequent solicited injection site reaction within 0-3 days following TENIVAC® was pain, reported in 78.3% of study participants 11-59 years of age and 35.3% of participants ≥60 years of age.
- The most frequent solicited systemic reaction within 0-3 days following TENIVAC® was headache, reported in 17.9% of participants, overall.
- Other common (≥10%) solicited adverse reactions within 0-3 days following TENIVAC® were injection site redness, injection site swelling, malaise, muscle weakness, and pain in joints. [11].

#### 2. STUDY OBJECTIVES

### 2.1. Primary Objective

• To evaluate the safety and tolerability of VIS649 in healthy subjects.

## 2.2. Secondary Objectives

- To characterize the PK profile of VIS649
- To evaluate the effect of ethnicity on the pharmacokinetic profile of a single intravenously (IV) dose of VIS649 in healthy Japanese and non-Japanese subjects
- To characterize the levels of anti-drug antibodies
- To characterize the effect of VIS649 on PD parameters including:
  - o changes in serum total IgA, IgG and IgM concentrations and time to recovery
  - o changes in circulating lymphocyte populations in cohorts 1-4 only (this assessment will be done for all lymphocytes, and also for lymphocyte subsets that are noted to show changes from baseline)
  - o assess ADA status impact on VIS649 PK parameters



#### 3. OVERALL DESIGN AND PLAN OF THE STUDY

#### 3.1. Overview

This is a Phase 1, randomized, placebo-controlled, double-blind, single ascending dose study to investigate the safety, tolerability, PK/PD of the IV administration of VIS649 in healthy subjects.

The study will be conducted in five sequential dosing cohorts. Cohorts 1-4 will enroll 9 subjects per cohort. Cohorts 1-4 will enroll 4 Japanese subjects and will be randomized to VIS649 or placebo in a ratio of 7:2 (7 active, 2 placebo). No more than one Japanese subject per cohort may be randomized to receive placebo. The fifth cohort will enroll up to 15 subjects with targeted but non-mandatory enrollment of up to 5 Japanese subjects. The subjects in cohort 5 will be randomized to VIS649 or placebo in a ratio of 10:5 (10 active, 5 placebo). No more than two Japanese subjects may be randomized to receive placebo in cohort 5.

The study is comprised of:

- A Screening Visit up to 28 days before dosing
- An in-house stay for approximately 2-3 days, with admission to the study center on Day -1, dosing on Day 1, and discharge in the morning of Day 2
- A post-administration period of 16 weeks
- Outpatient visits, on Day 3 (+1 day), 7 (± 1 day), 14, 21, 28, 31 (± 1 day) (cohort 5 only), 35, 42, 49 (cohorts 1-4 only), 56, 70, 84 and 98 (for all visits not otherwise specified, ± 3 days)
- A final Follow-up visit on Day 112 (± 3 days); Two additional follow-up visits may occur, at Weeks 20 and 24 post-dosing, if serum immunoglobulins have not returned to >lower limits of normal by the Week 16 (Day 112) visit, or if emerging trial data suggest a value of later follow-up (i.e., for detection of ADA responses).

The total duration of the clinical study per subject will be up to approximately 20 weeks (5 months), including the Screening period with the possibility of duration extending to 28 weeks (7 months) if follow-ups visits are required.

Potential subjects will be carefully screened for eligibility prior to study enrollment. Randomization and blinding will occur according to a core randomization list administered by the site's unblinded pharmacist. Back-up subjects who are not randomized into the cohort, but otherwise meet eligibility, may be re-screened after discussion among the Principal Investigator, Medical Monitor, and the Sponsor.

Eligible subjects will report to the Clinical Pharmacology Unit (CPU) at study check-in (Day -1) and will be required to stay in the CPU until Day 2 (24 hours post infusion). On Day 1, a single dose of VIS649 or placebo will be administered intravenously in the morning after a light meal (as per the clinical unit standard). Pharmacokinetics sampling will occur on Day 1 starting with a collection prior to the start of infusion, end of infusion, and at 2 hours, 8 hours and 24 hours post end of infusion. Pharmacokinetics samples will be collected on Days 1-3, 7, 14, 28, 42, 56, 70, and 112. Pharmacodynamics sampling (serum immunoglobulin levels, lymphocytes and sub Ig types) will occur as outlined in the Schedule of Assessments (see Table 10).



The initial cohort will be dosed with 0.5 mg/kg of VIS649. Escalation to next dosing level (2.0 mg/kg) will occur after review of blinded safety data through Day 14 by the Safety Monitoring Committee (SMC) comprised of the Principal Investigator, an independent Medical Monitor, and the Sponsor. Cohort 3 was reviewed after Day 56 data was collected to commence enrollment in cohort 4. Assessment of safety will be determined by evaluation of:

- Vital sign measurements
- Physical examinations
- Hematology, chemistry, and urinalysis laboratory testing
- 12-lead electrocardiograms (ECG)
- Adverse events, and
- Serum immunoglobulin levels

12 Mar 2019

Pharmacokinetic data will not be available for dose escalation decision making. Pharmacokinetic data will be reviewed in a blinded fashion after each cohort is available, and may result in a dose adjustment for subsequent cohorts. Any adjustments will be reviewed and approved by the Principal Investigator, Medical Monitor, and the Sponsor.

If dose escalation is stopped based on available blinded safety data, the current dose level will be considered as the minimum intolerable dose (MID). The dose just below the MID will be regarded as the maximum tolerated dose (MTD). If the dose escalation is stopped due to reaching exposure limit without dose limiting safety findings, the MTD will not be determined. Dose de-escalation may occur in additional cohorts, to further refine clinically relevant dose levels.

Stopping rules are described in Section 3.4.

Procedures related to the clinical study are detailed in the Schedule of Assessments (see Table 10).

Doses will be administered intravenously to subjects in approximately 5 dose cohorts (see Table 2). Cohorts are planned as follows:

**Table 2** Cohorts and Dose Administration

| Cohorts | Number of Subjects | Treatment |
|----------|--------------------|-------------------------------|
| Cohort 1 | N=7 | VIS649 0.5 mg/kg <sup>1</sup> |
| Conort 1 | N=2 | Placebo |
| Cohort 2 | N=7 | VIS649 2.0 mg/kg <sup>2</sup> |
| Conort 2 | N=2 | Placebo |
| Cohort 2 | N=7 | VIS649 6.0 mg/kg <sup>2</sup> |
| Cohort 3 | N=2 | Placebo |
| Cohort 4 | N=7 | VIS649 12 mg/kg |
| Conort 4 | N=2 | Placebo |
| Cohort 5 | N=10 | VIS649 6.0 mg/kg plus vaccine |
| Conort 3 | N=5 | Placebo plus vaccine |

<sup>&</sup>lt;sup>1</sup> After all subjects have completed assessments through Day 14, blinded safety data will be reviewed and a dose escalation decision for the subsequent cohort will be made by the SMC. If dose escalation is stopped, dose de-escalation may occur in additional cohorts, to further refine clinically relevant dose levels.

Please refer to Table 10 for a detailed list of procedures performed on each study day and visit.

<sup>&</sup>lt;sup>2</sup> After all subjects have completed assessments through Day 28, blinded safety data will be reviewed and a dose escalation decision for the subsequent cohort will be made by the SMC. If dose escalation is stopped, dose de-escalation may occur in additional cohorts, to further refine clinically relevant dose levels.

Figure 1 Study Flow Chart – Single Ascending Dose Design



#### 3.2. Endpoints

#### 3.2.1. Primary Endpoint

- Safety Endpoint
  - The proportion of subjects with AEs and serious adverse events (SAEs) following administration of VIS649; safety will be assessed from the time of study drug administration to the end-of-study participation.
- The following safety variables will be collected and recorded at regular intervals during the study:
  - Adverse event assessments
  - Clinical laboratory tests (hematology, clinical chemistry and urinalysis)
  - Vital signs (sitting BP, pulse, body temperature and respiratory rate [RR])
  - 12-lead ECG
  - Adjunctive procedures
  - Physical examination

#### 3.2.2. Secondary Endpoints

• Characterization of anti-drug antibodies (ADA) levels

#### 3.2.2.1. Pharmacokinetics Endpoints

The following PK parameters for VIS649 will be determined, as appropriate:

- C<sub>max</sub>: Maximum serum VIS649 concentration determined directly from the concentration-time profile
- T<sub>max</sub>: Time of maximum serum VIS649 concentration determined directly from the concentration-time profile
- AUC<sub>0-inf</sub>: Area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time
- AUC<sub>0-112d</sub>: Area under the concentration-time curve from pre-dose (time 0) to the concentration on Day 112
- AUC<sub>0-last</sub>: Area under the concentration-time curve from pre-dose (time 0) to the last quantifiable concentration

- t<sub>1/2</sub>: Apparent terminal elimination half-life
- Vd: Apparent volume of distribution
- CL: Apparent clearance

### 3.2.2.2. Pharmacodynamics Endpoints

- Changes in total serum IgG, IgA and IgM concentrations and time to recovery
- Changes in circulating lymphocyte populations in cohorts 1-4 only (this assessment will be done for all lymphocytes, and also for lymphocyte subsets that are noted to show changes from baseline).



#### 3.3. Justification of the Study Design

This study evaluates the safety, tolerability, and PK/PD of ascending single doses of VIS649 administered as an IV infusion. The design is standard and is considered appropriate to meet the objectives of the study.

A double-blind, placebo-controlled study is appropriate and standard for a single ascending dose study. This design will minimize bias and provide reference data (i.e., data from placebo-treated subjects) which will aid in the interpretation of results. The SMC will review available blinded safety, tolerability, and Ig level data after each cohort to confirm whether it is safe to proceed with the next planned dose, whether the dose escalation should be stopped or if the dose should be lowered, repeated, or titrated in the subsequent cohort.

The safety assessments for the study are accepted measures for ensuring safety of subjects during a clinical trial. The PK sampling schedule is considered appropriate given the information available. The rationale for dose selection is discussed in Section 5.3.

#### 3.4. Stopping Criteria for the Clinical Study and Dose Escalation Criteria

If any of the dose limiting toxicities listed below are met, the relevant subject(s) data may be unblinded. If the toxicity is present in  $\geq 1$  subject randomized to active drug, then dose escalation will pause. Depending upon the nature of the event, a decision may be made to resume dosing, to proceed into the next cohort at a lower dose level, or to stop the study.

Based on safety criteria, the dose adjustment/stopping criteria are as follows:

- Adverse event stopping criteria:
  - Any AE of severe intensity and related causality
  - Any SAE of related causality
- Vital sign stopping criteria:
  - Symptomatic hypotension (systolic blood pressure [SBP] <85 mmHg). If symptomatic hypotension that is related to the study drug is observed during the study, then a minimum of two repeat BP measurements should be obtained over a brief period. The mean of the three SBP measurements will be used to determine stopping criteria</p>
  - Tachycardia defined as heart rate >120 beats per minute (bpm) lasting longer than 30 minutes or with impaired consciousness
- Electrocardiogram stopping criteria:
  - QT interval
     (If a prolonged QTc interval is observed during the study, then a minimum of two repeat ECGs should be obtained over a brief period. The mean of the three ECGs will be used to determine stopping criteria.)
- Clinical laboratory stopping criteria:
  - Alanine aminotransferase (ALT)  $\geq 3$  times the upper limit of normal (ULN)
  - Aspartate aminotransferase (AST) ≥3 times the ULN
  - Serum creatinine >1.5 times the ULN
  - A decrease from baseline in hemoglobin concentration >3 g/dL
  - White blood cell count <1,500/mm<sup>3</sup>
  - Platelets < 50,000/mm<sup>3</sup>

| Visterra Inc. | Clinical Study Protocol |
|---------------|-------------------------|
| /IS649-101 | CONFIDENTIAL |

Visterra Inc.
# 4. STUDY POPULATION

The study population will consist of healthy Japanese and non-Japanese male and female volunteers. Subjects must be able to provide written informed consent and meet all the inclusion criteria and none of the exclusion criteria.

### 4.1. Number of Subjects

A total of 51 subjects may be enrolled in this clinical study. Cohorts 1-4 may have up to 36 subjects enrolled (a total of up to 16 Japanese subjects [up to 4 subjects each cohort] and up to 20 non-Japanese subjects [up to 5 subjects each cohort] [N=9 per dose cohort randomized to receive a single dose of VIS649 (N=7) or placebo (N=2)]). No more than 1 Japanese subject per cohort may be randomized to receive placebo in cohorts 1-4. Cohort 5 may have up to 15 subjects (N=15) with a targeted but non-mandatory enrollment of up to 5 Japanese subjects. Subjects in cohort 5 will be randomized to receive VIS649 (N=10) or placebo (N=5). In addition, all subjects in cohort 5 will receive TENIVAC® vaccine.

#### 4.2. Inclusion Criteria

Subjects who meet the following criteria will be considered eligible to participate in the clinical study:

- 1. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form prior to performing any of the Screening Visit procedures and be able to sign and date an appropriate Health Insurance Portability and Accountability Act (HIPAA) authorization form or subject privacy form, if appropriate.
- 2. Male and female subjects between 18 to 55 years of age, inclusive, at the Screening Visit.
- 3. For Japanese subjects: Subject is of Japanese descent as evidenced by verbal confirmation of familial heritage (a subject has all four Japanese grandparents born in Japan).
- 4. For non-Japanese subjects: Subjects must be of non-Asian descent, as evidenced by verbal confirmation that all four grandparents are non-Asian.
- 5. The following applies to female subjects:
  - Non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation]) for at least 6 months, or postmenopausal ≥ 1 year, or

Amendment 2, Version 3.0  12 Mar 2019

- Non-pregnant, non-lactating females of childbearing potential must report prior use (over the 28 days prior to dosing of study drug) of medically acceptable forms of birth control (hormonal contraception, abstinence, diaphragm with spermicide, condom with spermicide or intrauterine device, or partner with vasectomy), with agreement to continue to use a medically acceptable form of birth control (as described) through the end of their participation in the study. Alternatively, a reported history of abstinence beginning at least 28 days prior to study drug dosing, with agreement to continue abstinence through the end of their participation in the study are required. Females of childbearing potential must also have a negative serum human chorionic gonadotropin (hCG) pregnancy test at Screening and a negative urine hCG pregnancy test at baseline (Day -1). Female subjects must also agree not to donate eggs/bank eggs for the duration of their participation in the study.
- 6. For male, subject and/or his partner must use a highly effective form of contraception (i.e., double-barrier as described above, have had a vasectomy, or have a female partner of non-childbearing potential) or agree to abstinence following study drug dosing, through the end of the subject's participation in the study. Male subjects must also agree to not donate sperm for the duration of their participation in the study, following study drug dosing.
- 7. Screening laboratory values must meet the following criteria:
  - White blood cells  $3,000-12,000/\text{mm}^3$
  - Platelets  $>150,000/\text{mm}^3$
  - Hemoglobin >13 gm/dL for male and>11 gm/dL for female
  - Estimated glomerular filtration rate >80 mL/min/1.73 m<sup>2</sup> (using the Modification of Diet in Renal Disease study equation)
  - Serum creatinine <1.25x ULN
  - Blood Urea Nitrogen (BUN) ≤25mg/dL
  - Aspartate aminotransferase (AST) ≤50 U/L
  - Alanine aminotransferase (ALT) ≤67 U/L
  - Alkaline phosphatase ≤150 U/L
  - Total Bilirubin ≤1.4 mg/dL

unless patient has Gilbert Syndrome, in which case direct bilirubin must be within normal range

Amendment 2, Version 3.0  12 Mar 2019



- 8. Body mass index (BMI) between 18 and 32 kg/m<sup>2</sup>, inclusive, at the Screening Visit.
- 9. Healthy, determined by pre-study medical evaluation (medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations), as judged by the Principal Investigator.
- 10. Is willing and able to comply with study restrictions and to remain at the CPU for the in-patient duration of the study and return for all follow-up outpatient visits.
- 11. QTcF < 450 msec at Screening (may be repeated once).

#### 4.3. Exclusion Criteria

Subjects who meet one or more of the following criteria will not be considered eligible to participate in the clinical study:

- 1. Is participating in another clinical study of any investigational drug, device, or intervention or has received any investigational medication during the last 30 days or 5 half-lives, whichever is longer, before baseline (Day -1).
- 2. Subject is judged by the Principal Investigator or the Medical Monitor to be inappropriate for the study.
- 3. Subject has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, blood dyscrasias or other medical disorder, including psychiatric disorders, cirrhosis or malignancy. History of minor skin cancers (not including melanoma) or surgically treated, limited cervical carcinomas (i.e., carcinoma in situ) are not exclusionary.
- 4. Subject has a history or presence of proteinuria, chronic kidney disease, disease requiring immunosuppressive therapy (including systemic steroids), or is considered to be immunosuppressed for any other reason.
- 5. Previous receipt of antibody or biologic therapy whether licensed or investigational (immunoglobulin products, monoclonal antibodies or antibody fragments) within 30 days

Amendment 2, Version 3.0  12 Mar 2019

- prior to dosing or 5 half-lives within the dose of Investigational medicinal product (IMP), whichever is longer.
- History of a previous severe allergic reaction with generalized urticaria; angioedema or anaphylaxis.
- 7. History of severe allergic reaction (e.g. anaphylaxis) to a previous dose of TENIVAC®, or any other tetanus/diphtheria toxoid-containing vaccine, or any component of this vaccine.
- 8. History of an Arthus-type hypersensitivity reaction to tetanus vaccine in the past (a reaction characterized by severe pain, swelling, induration, edema and bruising, with onset typically 4 to 12 hours after vaccination).
- 9. History of having Guillain-Barre syndrome
- 10. Has received a tetanus vaccine in the past 5 years.
- 11. Blood pressure >160/100 mmHg or <90/50 mmHg (may be repeated once if abnormal), at the Screening visit and Day -1.
- 12. Known hypoglobulinemia disorder (i.e., common variable immunodeficiency), X-linked agammaglobulinemia, selective IgA deficiency, selective IgM deficiency).
- 13. History of pre-existing latent infections (e.g., tuberculosis) or any infection requiring hospitalization or treatment with antivirals or antibiotics, or vaccination within 30 days prior to administration of study medication.
- 14. Concomitant use of marketed or investigational systemic immunosuppressive or immunomodulatory medications (e.g., corticosteroids, methotrexate, azathioprine, etc. and/or biologics) is prohibited and require a washout period prior to Screening (30 days or 5 half-lives, whichever is longer).
- 15. Has received any prescription or non-prescription (over-the-counter [OTC]) medication during the last 30 days or 5 half-lives, whichever is longer, preceding baseline (Day -1), with the exception of acetaminophen, ibuprofen, hormonal contraceptives, topical medications, vitamins, and dietary or herbal remedies.
- 16. Subjects who consume more than 21 units of alcohol per week (7 days) or those who have a history of alcohol or drug/chemical abuse; one unit of alcohol is equivalent to eight ounces of beer, 4 ounces of wine, or one ounce of spirits.
- 17. Subject is a user or former user of nicotine-containing products (including but not limited to cigarettes, cigars, and chewing or dipping tobacco) who stopped use or consumption (i.e.,

smoking, chewing, or pinching) of these nicotine-containing products less than 3 months before study drug administration or is using or has used topical or oral nicotine preparations for smoking cessation within the past 90 days before study drug administration.

- 18. Subjects who consume greater than 500 mg of caffeine or xanthine-containing products per day (e.g., coffee, tea, soft drinks, energy drinks, or chocolate).
- 19. Subjects who refuse to abstain from alcohol, xanthine-containing or caffeine-containing foods or beverages from 48 hours prior to check-in on Day-1 through the end of the study.
- 20. Subjects with a positive urine drug (inclusive of marijuana), alcohol, or cotinine Screening test result at Screening and Day-1. The urine drug screen also screens for methylenedioxymethamphetamine, tricyclic antidepressants, oxycodone, and propoxyphene. If a subject tests positive on these extra 4 tests, inclusion of that subject into the study will be based on the Principal Investigator's judgment with consultation, as needed, with the Medical Monitor and the Sponsor.
- 21. Subjects with a positive hepatitis B surface antigen test or evidence of chronic hepatitis C virus infection at Screening (a negative HCV antibody assay at Screening is sufficient to rule-out chronic HCV infection for this study).
- 22. Subjects with a known history of a positive Human Immunodeficiency Virus (HIV) or a positive test result at Screening.
- 23. Subjects who have donated >500 mL or blood within 60 days prior to start of Screening.
- 24. The subject has donated any plasma within 7 days prior to baseline (Day -1).
- 25. Is an employee of the clinical research team (any Sponsor or research site employee), or has a family member who is an employee of these organizations.

# 4.4. Subject Withdrawal and Replacement

While subjects are encouraged to complete all study evaluations, they may withdraw from the study at any time and for any reason. Every effort will be made to determine why any subject withdraws from the study prematurely. All subjects who withdraw from the study with an ongoing AE must be followed until the event is resolved or deemed stable. If a subject withdraws prematurely after dosing, all data to be collected prior to discharge from the clinical site should be collected at the time of premature discontinuation or at the scheduled discharge. Subject participation may be terminated prior to completing the study and the reason recorded as follows:

#### 1. Adverse event

- 2. Protocol violation
- 3. Loss to follow-up
- 4. Subject withdrew consent at own request
- 5. Other

A genuine effort must be made to determine the reason(s) why a subject fails to return for the necessary visits or is discontinued from the study. If the subject is unreachable by telephone, a registered letter, at the minimum, should be sent to the subject requesting him/her to contact the clinic.

Subjects can be replaced, and a replacement randomization number will be generated. The same treatment will be allocated to the replacement subject.

# 4.5. Termination of the Clinical Study

If the Principal Investigator, the Sponsor, or the Medical Monitor becomes aware of conditions or events that suggest a possible hazard to subjects if the clinical study continues, then the clinical study may be terminated after appropriate consultation among the involved parties. The clinical study may be terminated at the Sponsor's discretion also in the absence of such a finding.

Conditions that may warrant termination of the clinical study include, but are not limited to:

- The discovery of an unexpected, relevant or unacceptable risk to the subjects enrolled in the clinical study;
- Failure to enroll subjects at the required rate;
- A decision of the Sponsor to suspend or discontinue development of the study drug.

Should the study be terminated and/or the site closed for whatever reason, all documentation pertaining to the study and VIS649 must be returned to the Sponsor. Any actions of PAREXEL required for assessing or maintaining subject safety will continue as required, despite termination of the study by the Sponsor.

#### 5. INVESTIGATIONAL MEDICINAL PRODUCT AND TOXOID VACCINATION

# 5.1. Identity of the Investigational Medicinal Products

The investigational products that will be used in this study are outlined in Table 3.

Table 3 Identity of Investigational Products

| Drug Name | Formulation | Strength | Route | Manufacturer |
|---|---|---|---|---|
| VIS649 | Solution<br>(to be diluted into a<br>final volume of<br>100 mL 0.9% NaCl) | 25 mg/mL | IV | Sponsor |
| Placebo | Solution | 0.9% NaCl | IV | To be sourced by PAREXEL |

IV: intravenous; NA: not applicable; NaCl: Sodium Chloride

Data source: Investigator Brochure

# 5.2. Tetanus/Diphtheria Toxoid Vaccine (TENIVAC®)

The tetanus/diphtheria toxoid vaccine that will be used in this study is outlined in Table 4.

Table 4 Tetanus/Diphtheria Toxoid Vaccine

| Vaccine Name | Formulation | Strength | Route | Manufacturer |
|--------------|-------------|----------|-------|--------------|
| TENIVAC® | Solution | NA | IM | Sanofi |

IM: Intramuscular; IV: intravenous; NA: not applicable; NaCl: Sodium Chloride

# 5.3. Rationale for Starting Dose and Dose Escalation

VIS649 will be administered at a first-in-human starting dose of 0.5 mg/kg IV to healthy volunteers. The starting dose was selected upon consideration of the VIS649 target and mechanism of action, *in-vitro/in-vivo* toxicology data, the NOAEL observed in the pivotal toxicology study in cynomolgus monkeys, and estimations derived from a PK/PD model of the pharmacologically active dose in humans. In each dosing cohort, two subjects (one receiving placebo, the other receiving VIS649) will be dosed 24 hours before others in the respective cohort, to provide a sentinel function should unanticipated adverse reactions occur at any dose level.

The cynomolgus monkey is considered a relevant species for evaluation of VIS649 toxicity due to similarity in B-cell biology, 99% sequence homology between cynomolgus and human APRIL, and similar binding affinity of VIS649 to cynomolgus and human APRIL (within ~2-fold). The effects of multiple doses of VIS649 were evaluated in a GLP toxicology study in

healthy cynomolgus monkeys at 25, 50, and 100 mg/kg IV once weekly over 28 days. VIS649 was well tolerated in cynomolgus monkeys with no VIS649-related clinical findings up to 100 mg/kg; the NOAEL from this study was 100 mg/kg.

A maximum recommended starting dose of 5 mg/kg was identified by considering the NOAEL of 100 mg/kg in cynomolgus monkeys, which translates to a human equivalent dose of 100 mg/kg for monoclonal antibody therapeutics. Applying a safety factor of 2X that accounts for the measured affinity difference of VIS649 for monkey and human APRIL, and an additional 10X safety factor to account for potential interspecies differences and other unknowns arrives at a NOAEL justified starting dose of 5 mg/kg, which is expected to be well tolerated in humans based on cynomolgus monkey studies.





The minimum pharmacologically active dose of 0.5 mg/kg was selected as the starting dose for evaluation in healthy volunteers; this is 10-fold lower than the maximum recommended starting dose based on the NOAEL. Doses from 0.5 to 12 mg/kg will be evaluated in single dose escalation in four cohorts, with a final cohort to receive a dose of 6.0 mg/kg. Dose escalations will not exceed a 4-fold increase. The safety margins for targeted clinical doses are provided in Table 5.



# 5.4. Supply, Packaging, Labeling and Storage

Investigational medicinal products will be packaged and labeled according to applicable local and regulatory requirements.



All supplies of study drug VIS649 must be stored between≥2°C and ≤8°C and protected from light. The study drug VIS649 will be stored in a securely locked area, accessible to authorized persons only.

### 5.5. Drug Accountability, Dispensing and Destruction

The Principal Investigator or designee is responsible for maintaining accurate accountability records of the study drug and TENIVAC® vaccine throughout the clinical study. The drug accountability log includes information such as, randomization number, amount dispensed and amount returned to the pharmacy (if any). Products returned to the pharmacy will be stored under the same conditions as products not yet dispensed. The returned products should be marked as 'returned' and kept separate from the products not yet dispensed.

All dispensing and accountability records will be available for Sponsor review. When the Study Monitor visits PAREXEL, he/she will reconcile the drug accountability log with the products stored in the PAREXEL pharmacy.

The PAREXEL pharmacist (or designee under the direction of the pharmacist) will dispense study drug and TENIVAC® vaccine in a blinded manner for each subject according to the protocol, randomization list and pharmacy manual, if applicable.

After receiving Sponsor approval in writing, PAREXEL is responsible for returning all unused or partially used study drug to the Sponsor or designated third party or for preparing the study drug for destruction via carbonization.

# 5.6. Subject Identification and Randomization

# **5.6.1.** Screening Numbers

All screened subjects are assigned a unique 3-digit subject identification (SID) number (001 - 999). The SID numbers identify subjects from time of Screening until time of randomization. Enrolled subjects who drop out of the clinical study before randomization will retain their SID numbers.

### **5.6.2.** Randomization Numbers

Prior to dosing on Day 1, eligible subjects will be assigned a randomization number in accordance with the randomization code generated by PAREXEL International. The randomization code will be maintained in a room with restricted access to pharmacy personnel only. The randomization code will include 4-digit subject numbers Cohort and randomization numbers are listed in Table 6.

 Table 6
 Randomization Numbers and Treatment Assignment

| Dose<br>Group | Randomization<br>Numbers | Replacement<br>Numbers | Treatment Assignment | |
|---|---|---|---|---|
| Cohort 1 | | | 0.5 mg/kg VIS649 (N=7) | Placebo (N=2) |
| Cohort 2 | | | 2.0 mg/kg VIS649 (N=7) | Placebo (N=2) |
| Cohort 3 | | | 6.0 mg/kg VIS649 (N=7) | Placebo (N=2) |
| Cohort 4 | | | 12 mg/kg VIS649 (N=7) | Placebo (N=2) |
| Cohort 5 | | | 6.0 mg/kg VIS649 (N=10) | Placebo (N=5) |

Once a randomization number has been allocated to one subject, it may not be assigned to another subject. If subjects withdrawn prematurely from the study and are replaced under the direction of the Sponsor, then a replacement randomization number will be assigned. A replacement randomization code will be generated such that replacement subjects are assigned to the same treatment as the discontinued subjects. The replacement randomization code will differ only in randomization numbers, which will be 4-digit numbers

No more than one Japanese subject per cohort may be randomized to receive placebo in cohorts 1-4.

The full randomization code will be broken for purposes of final data analysis and reporting of final TLFs after final database lock. This will occur once all final data have been entered into the database and all data queries have been resolved, coding is complete, the assignment of subjects to the analysis sets has been completed and the database has been locked.

# 5.7. Administration of Investigational Medicinal Products

The amount of VIS649 will be calculated on a per subject weight basis and administered diluted in 100 mL of 0.9 % sodium chloride. Subject weight will be captured after admission to the research unit (Day -1) and will be used by the pharmacy staff for subject-specific dose calculation. VIS649 will be administered intravenously using a volumetric pump and through a 0.22µm in line IV filter at a rate of 100 mL/hr over the course of one hour. A saline flush is performed after the infusion is complete to ensure that any drug product remaining in the infusion line is administered. Placebo will be 100 mL of 0.9% sodium chloride administered IV in an identical manner.

For cohort 5 participants, on Day -1, a single dose of VIS649 or placebo will be administered intravenously in one arm and on Day 28, a single dose of tetanus/diphtheria vaccine will be injected intramuscularly into the opposite arm.

Refer to the pharmacy manual for specific details on storage, handling, and preparation information.

# **5.8.** Compliance

Dosing will be performed by trained, qualified personnel designated by the Principal Investigator. The date, time and volume of the administered dose will be documented. Comments will be recorded if there are any deviations from the planned dosing procedures.

# 5.9. Blinding and Breaking the Blind

The clinical study will be performed in a double-blind manner, for clinical research unit staff interacting with study participants, with the exception of the persons involved in the preparation of the IMPs. These persons will not be involved in any other study activities.

Prior to scheduled unblinding as described below, the study blind should not be broken except in a medical emergency (where knowledge of the study drug administered would affect the treatment of the emergency). The decision to break the blind will be made on a case-by-case basis, at the discretion of the Principal Investigator in collaboration with the Sponsor/Medical Monitor. The applicable Standard operating procedure (SOP) will be followed for blind breaking procedures.

As participants in each dosing cohort complete their Week 16 visit, data clean-up and soft-lock will be performed for cohorts 1-4 only, in order to allow interim assessments of blinded data. PK/PD analysts will have access to unblinded data at all times, but those individuals will not be involved in study participant interactions. Summaries of treatment specific PD responses (principally, individual immunoglobulin levels over time and group mean, median, minimum and maximum parameters by treatment assignments) will be prepared and shared with the Sponsor, in a manner that does not unblind individual patient treatment assignments. A registry of dummy subject identifiers will be created. A physician who is not involved in the study will review Ig results to maintain the blind for the Principal Investigator.

#### 5.10. Prior and Concomitant Medications

Any medicinal product, prescribed or OTC, including herbal and other nontraditional remedies, is considered a concomitant medication. Prior and concomitant medication use will be recorded for the 30 days prior to the Screening Visit until the End-of-study Visit. Prior and concomitant medication use is not permitted during the last 30 days or 5 half-lives, whichever is longer, preceding baseline (Day -1) until end-of-study (including prescription or non-prescription [over-the-counter]) medication, except for acetaminophen, ibuprofen, hormonal contraceptives, topical medications, vitamins, dietary or herbal remedies). However, concomitant medication use may be warranted for the treatment of AEs. The use of concomitant medications to treat AEs should be discussed between the Principal Investigator and the Medical Monitor.

# 5.11. Treatment of Overdose

Standard symptomatic support measures should be used in the case of excessive pharmacological effects or overdose. No antidotes are available.

# 6. MEASUREMENTS AND METHODS OF ASSESSMENT

For timing of assessments, refer to the Schedule of Assessments (Table 10).

A Safety Management Plan will be signed between the Sponsor and PAREXEL.

# 6.1. Medical History, Demographic and Other Baseline Information

The medical history comprises:

- General medical history
- Medication history
- Reproductive history

The following demographic information will be recorded:

- Age
- Ethnicity: Japanese or non-Japanese
- Race: White, Black, Hispanic/Latino, American Indian/Alaska native, Asian, Pacific Islander
- Height, without shoes (cm)
- Body weight, without shoes (kg)
- BMI  $(kg/m^2)$

Other baseline characteristics will be recorded as follows:

- History of drug abuse
- History of alcohol abuse
- Smoking history
- History of caffeine use (or other stimulating beverages)
- History of blood or plasma donation
- Date of most recent tetanus/diphtheria toxoid vaccination

# **6.2.** Safety Variables

#### **6.2.1.** Adverse Events

Adverse event reporting will begin for each subject from baseline (Day -1) and will continue until the End-of-study Visit.

# **6.2.1.1.** Definitions

#### **6.2.1.1.1. Definition of Adverse Event**

Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

Other untoward events occurring in the framework of a clinical study will be recorded as AEs, e.g. those occurring during treatment-free periods (including post-dosing periods), in association with study-related procedures and assessments, or under placebo. For study drugs, lack of efficacy may be an expected potential outcome and should not be reported as an AE unless the event is unusual in some way, e.g., greater in severity.

Concomitant illnesses, which existed prior to entry into the clinical study, will not be considered AEs unless they worsen during the treatment period. Pre-existing conditions will be recorded as part of the subject's medical history.

### **6.2.1.1.2. Definition of Serious Adverse Event**

An SAE is defined as any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening; this means that the subject was at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe
- Requires in-patient hospitalization or prolongation in existing hospitalization
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
- Is a congenital anomaly/birth defect, or
- Is another important medical event (see below)

Important medical events that do not result in death, are not life-threatening or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or in a physician's office, blood dyscrasias or seizures that do not result in in-patient hospitalization, and the development of drug dependency or drug abuse.

A distinction should be drawn between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria above. For example, a mild degree of gastrointestinal bleeding requiring an overnight hospitalization for monitoring purposes would be considered an SAE, but is not necessarily severe. Similarly, an AE that is severe in intensity is not necessarily an SAE. For example, alopecia may be assessed as severe in intensity but would not be considered an SAE.

Medical and scientific judgment should be exercised in deciding if an AE is serious and if expedited reporting is appropriate.

# **6.2.1.1.3.** Adverse Events of Special Interest

An adverse event of special interest (serious or non-serious) is one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Principal Investigator to the Sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it. Depending on the nature of the event, rapid communication by the Sponsor to other parties might also be warranted.

Examples of these are all AEs of

- Infusion reactions: Fever, chills, rigors, nausea, vomiting, pain, headache, dizziness, shortness of breath, bronchospasm, hypotension, hypertension, pruritus, rash, urticaria, angioedema, diarrhea, tachycardia, and chest pain
- Delayed allergic reactions: Serum sickness (i.e., urticaria, fever, general glandular enlargement, joint pains)
- General: Injection site reaction
- Any documented infection

# **6.2.1.2.** Recording of Adverse Events

Adverse events should be collected and recorded for each subject from the baseline (Day -1) until the end of their participation in the study, i.e. the subject has discontinued or completed the study.

Adverse events may be volunteered spontaneously by the subject, or discovered by the study staff during physical examinations or by asking an open, non-leading question such as 'How have you been feeling since you were last asked?' All AEs and any required remedial action will be recorded. The nature of AE, date (and time, if known) of AE onset, date (and time, if known) of AE outcome to date, severity and action taken of the AE will be documented together with the Principal Investigator's assessment of the seriousness of the AE and causal relationship to study drug and/or study procedure.

All AEs should be recorded individually in the subject's own words (verbatim) unless, in the opinion of the Principal Investigator, the AEs constitute components of a recognized condition, disease or syndrome. In the latter case, the condition, disease or syndrome should be named rather than each individual symptom. The AEs will subsequently be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 21.0 or higher).

# **6.2.1.3.** Assessment of Adverse Events

Each AE will be assessed by the Principal Investigator with regard to the categories discussed in the following sections.

#### **6.2.1.3.1.** Intensity

The Principal Investigator will assess all AEs for severity in accordance with the following standard ratings.

- Mild: Ordinarily transient symptoms, does not influence performance of subject's daily activities. Treatment is not ordinarily indicated.
- Moderate: Marked symptoms, sufficient to make the subject uncomfortable. Moderate influence on performance of subject's daily activities. Treatment may be necessary.
- Severe: Symptoms cause considerable discomfort. Substantial influence on subject's daily activities. May be unable to continue in the study and treatment may be necessary.

When changes in the intensity of an AE occur more frequently than once a day, the maximum intensity for the event should be noted for that day. Any change in severity of signs and

symptoms over a number of days will be captured by recording a new AE, with the amended severity grade, and the date (and time, if known) of the change.

# **6.2.1.3.2.** Causality

The Principal Investigator will assess the causality/relationship between the study drug and the AE. One of the categories described in Table 7 should be selected based on medical judgment, considering the definitions below and all contributing factors.

Table 7 Assessment of Relationship of Adverse Events to Investigational Product/and or Vaccine

| Related | A clinical event, including laboratory test abnormality, occurs in a plausible time relationship to treatment administration, and which concurrent disease or other drugs or chemicals cannot explain. The response to withdrawal of the treatment (de-challenge*) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory re-challenge† procedure if necessary. |
|---|---|
| Probably related | A clinical event, including laboratory test abnormality, with a reasonable time sequence to administration of the treatment, unlikely to be attributed to concurrent disease or other drugs or chemicals, and which follows a clinically reasonable response on withdrawal (de-challenge). Re-challenge information is not required to fulfil this definition. |
| Possibly related | A clinical event, including laboratory test abnormality, with a reasonable time sequence to administration of the treatment, but which could also be explained by concurrent disease or other drugs or chemicals. Information on treatment withdrawal may be lacking or unclear. |
| Unlikely to be related | A clinical event, including laboratory test abnormality, with a temporal relationship to treatment administration which makes a causal relationship improbable, and in which other drugs, chemicals or underlying disease provide plausible explanations. |
| Unrelated | A clinical event, including laboratory test abnormality, with little or no temporal relationship with treatment administration. May have negative de-challenge and re-challenge information. Typically explained by extraneous factors (e.g., concomitant disease, environmental factors or other drugs or chemicals). |

<sup>\*</sup>De-challenge is when a drug suspected of causing an AE is discontinued. If the symptoms of the AE disappear partially or completely, within a reasonable time from drug discontinuation, this is termed a positive de-challenge. If the symptoms continue despite withdrawal of the drug, this is termed a negative de-challenge. Note that there are exceptions when an AE does not disappear upon discontinuation of the drug, yet drug-relatedness clearly exists (for example, as in bone marrow suppression, fixed drug eruptions, or tardive dyskinesia).

#### **6.2.1.3.3.** Seriousness

Severity is a measure of intensity whereas seriousness is defined by the criteria in Section 6.2.1.1.2.

# **6.2.1.4.** Reporting of Serious Adverse Events

The Principal Investigator will review each SAE and evaluate the intensity and the causal relationship of the event to study drug. All SAEs will be recorded from signing of the ICD until

<sup>†</sup>Re-challenge is when a drug suspected of causing an AE in a specific subject in the past is re-administered to that subject. If the AE recurs upon exposure, this is termed a positive re-challenge. If the AE does not recur, this is termed a negative re-challenge.

the End-of-study Visit. Serious AEs occurring after the End-of-study Visit and coming to the attention of the Principal Investigator must be reported only if there is (in the opinion of the Principal Investigator) reasonable causal relationship with the study drug.

The Principal Investigator is responsible for providing notification to the Clinical Research Organization (CRO)/Sponsor of any SAE, whether deemed IMP-related or not, that a subject experiences during their participation in study within 24 hours of becoming aware of the event.

As a minimum requirement, the initial notification should provide the following information:

- Study number
- Patient number
- Sex
- Date of birth
- Name of Principal Investigator and full clinical site address
- Details of SAE
- Criterion for classification as 'serious'
- Study drug name, or code if unblinded, and treatment start date
- Date of SAE onset
- Causality assessment (if sufficient information is available to make this classification)

The CRO/Sponsor will request clarification of omitted or discrepant information from the initial notification. The Principal Investigator or an authorized delegate is responsible for emailing or faxing the requested information to the CRO/Sponsor within 24 hours of the request.

Initial reports of SAEs must be followed later with detailed descriptions, including clear photocopies of other documents as necessary (e.g. hospital reports, consultant reports, autopsy reports), with the subject's personal identifiers removed. All relevant information obtained by the Principal Investigator through review of these documents will be recorded and faxed to the Sponsor within 24 hours of receipt of the information. If a new SAE Report Form is faxed, then the Principal Investigator must sign and date the form. The CRO/Sponsor may also request additional information on the SAE, which the Principal Investigator or an authorized delegate must fax to the Sponsor within 24 hours of the request.

# **Serious Adverse Event Reporting:**

PAREXEL Safety Services



All AEs experienced by a subject, irrespective of the suspected causality, will be monitored until the event has resolved, until any abnormal laboratory values have returned to baseline or stabilized at a level acceptable to the Principal Investigator and Medical Monitor, until there is a satisfactory explanation for the changes observed or until the subject is lost to follow-up.

# **6.2.1.6. Pregnancy**

The Sponsor has a responsibility to monitor the outcome of all pregnancies reported during the clinical study.

Pregnancy alone is not regarded as an AE unless there is a suspicion that the study drug may have interfered with the effectiveness of a contraceptive medication. Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions (see below). Hospitalization for normal delivery of a healthy newborn should not be considered an SAE.

Each pregnancy must be reported by the Principal Investigator to the Sponsor within 24 hours after becoming aware of the pregnancy. The Principal Investigator must follow-up and document the course and the outcome of all pregnancies even if the subject was withdrawn from the clinical study or if the clinical study has finished.

All outcomes of pregnancy must be reported by the Principal Investigator to the Sponsor on the pregnancy outcome report form within 24 to 48 hours after he/she has gained knowledge of the normal delivery or elective abortion.

Any SAE that occurs during pregnancy must be recorded on the SAE Report Form (e.g., maternal serious complications, therapeutic abortion, ectopic pregnancy, stillbirth, neonatal death, congenital anomaly, birth defect) and reported within 24 hours in accordance with the procedure for reporting SAEs.

# **6.2.2.** Clinical Laboratory Assessments

Samples for clinical laboratory assessments will be collected at the time points detailed in the Schedule of Assessments (see Table 10). Clinical laboratory tests will be performed by the laboratories mentioned in the List of Study Staff of this clinical study protocol. Samples will be collected in appropriate tubes and handled according to standard procedures of the applicable laboratory.

Table 8 lists the biochemistry, hematology and urinalysis tests that will be performed by the local laboratory for safety blood samples.

| Table 8 | Clinical Laboratory A | ssessments |
|---------|-----------------------|------------|
|---------|-----------------------|------------|

| Hematology | |
|---|---|
| White blood cell (WBC) count | Neutrophils (percentage and absolute count) |
| Red blood cell (RBC) count | Lymphocytes (percentage and absolute count) |
| Hemoglobin (Hb) | Monocytes (percentage and absolute count) |
| Hematocrit (HCT) | Eosinophils (percentage and absolute count) |
| Mean corpuscular volume (MCV) | Basophils (percentage and absolute count) |
| Mean corpuscular hemoglobin (MCH) | Platelet count |
| Mean corpuscular hemoglobin concentration (MCHC) | RBC distribution width |
| Coagulation | |
| Prothrombin time (PT) | International Normalized Ratio (INR) |
| Activated partial thromboplastin time (aPTT) | |
| Clinical Chemistry | |
| Alanine aminotransferase (ALT) | Glucose |
| Albumin | Lactate dehydrogenase (LDH) |
| Alkaline phosphatase (ALP) | Phosphorus |
| Aspartate aminotransferase (AST) | Potassium |
| Blood urea nitrogen (BUN) | Sodium |
| Calcium | Total bilirubin |
| Chloride | Total protein |
| Cholesterol | Triglycerides |
| Creatinine | Uric acid |
| Gamma glutamyl transferase (GGT) | |
| SH (Screening Visit only; all female subjects) | |
| J <b>rinalysis</b> | |
| Bilirubin | Blood |
| Glucose | pH and specific gravity |
| Ketones | Protein |
| Leukocytes | Urobilinogen |
| Nitrite | |
| Microscopic (only for abnormal urine stick test findings) | |
| Serology | |
| Human immunodeficiency virus (HIV) | Hepatitis C virus antibody (anti-HCV) |
| Types 1 and 2) antibodies | Tetanus/diphtheria serology |
| Hepatitis B surface antigen (HBsAg) | |
| Urine Drug Screening and Cotinine Test | |
| Amphetamines | Cocaine |
| Barbiturates | Opiates |
| Benzodiazepines | Phencyclidine |
| Cannabinoids | Cotinine |
| Urinary creatinine (to exclude dilution effect) | Ethanol |
| Pregnancy Testing | |
| Serum/urine human beta chorionic gonadotrophin (women | en of childbearing notential only) |

Abnormal laboratory results should be recorded as AEs (e.g., Principal Investigator judgment or outside the specific reference range).

Any value outside the normal range will be flagged for the attention of the Principal Investigator or designee at the site. The Principal Investigator or designee will indicate whether or not the value is of clinical significance. If the result of any test (or repeat test, if done) from the samples taken during the Screening period is indicated as clinically significant, the subject will not be allowed into the study without permission of the Medical Monitor. Additional testing during the study may be done if medically indicated. If a clinically significant abnormality is found in the samples taken after dosing, during the study, and/or at the End-of-study Visit, it should be recorded as an AE and the subject will be followed until the test(s) has (have) normalized or stabilized, at the discretion of the Principal Investigator.

# 6.2.2.1. Anti-drug Antibody Response

The serum samples to measure the presence of ADA will be collected on Days 1, Week 4,8,16 and if required Weeks 20 and 24. The presence or absence of ADA will be determined in the serum samples using validated bioanalytical methods. Blood samples for ADA analysis will be collected up to Week 16 from all subjects. Samples for anti-VIS649 antibody titers and neutralizing capabilities will be drawn according to the Schedule of Assessments (see Table 10). Further procedures for sample collection, shipment, processing and storage will be described in the Laboratory Manual.

# 6.2.3. Vital Signs

Vital signs will be assessed at the time points detailed in the Schedule of Assessments (see Table 10). The following vital signs will be measured:

- Blood pressure (systolic and diastolic [mmHg])
- Pulse (bpm)
- Respiratory rate (breaths per minute)
- Temperature

Blood pressure and pulse recordings will be made after the subject has been in a seated or supine position and at rest > 5 minutes.

### 6.2.4. Standard 12-lead Electrocardiograms

Standard safety 12-lead ECGs will be performed at the time points detailed in the Schedule of Assessments (see Table 10).

The 12-lead ECGs will be performed after the subject has been resting supine for≥ 5 minutes. The ECG will include all 12 standard leads and a Lead II rhythm strip on the bottom of the tracing. The ECG will be recorded at a paper speed of 25 mm/sec. The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval and QTc interval (QTcF).

All ECGs must be evaluated by a qualified physician or physician's assistant for the presence of abnormalities.

### 6.2.5. Physical Examinations

Physical examinations will be performed at the time points detailed in the Schedule of Assessments (see Table 10).

Full physical examination:

An assessment of general appearance and a review of systems (dermatologic, head, eyes, ears, nose, mouth/throat/neck, thyroid, lymph nodes, respiratory, cardiovascular, gastrointestinal, extremities, musculoskeletal, neurologic and psychiatric systems).

Brief physical examination:

An assessment of the general appearance, skin, cardiovascular system, respiratory system and abdomen.

The brief physical examination may be extended to a full physical examination if considered necessary by the Principal Investigator. Other evaluations may be performed as deemed necessary by the Principal Investigator. This will be commented upon in the clinical study report (CSR), if performed.

#### 6.3. Pharmacokinetics Variables

### **6.3.1.** Blood Sample Collection

Blood for the analysis of VIS649 will be collected at the time points detailed in the Schedule of Assessments (see Table 10).

12 Mar 2019

Blood sample collection, processing and shipping details will be outlined in a separate laboratory manual. In brief, PK sampling will occur on Day 1 starting with a collection prior to the start of infusion, at the end of infusion (60 minutes) and at 2 hours, 8 hours and 24 hours post end of infusion. Pharmacokinetics samples will also be drawn on Days 3, 7, 14, 28, 42, 56, 70, and 112. Serum samples for determination of the concentration of VIS649 will be analyzed under the responsibility of the Sponsor. Further procedures for sample collection, shipment, processing, and storage will be described in the Laboratory Manual.

# 6.4. Pharmacodynamics Variables



Samples for PD parameters will be collected at the time points detailed in the Schedule of Assessments (see Table 10). Further procedures for sample collection, shipment, processing, and storage will be described in the Laboratory Manual.

#### 6.5. Total Amount of Blood

The approximate volume of blood (440.5 mL) planned for collection from each subject over the course of the entire study (from the Screening Visit to the End-of-study Visit, but not including repeat or additional tests ordered by the Principal Investigator) presents no undue risk to the subjects.

For all subjects enrolled, the approximate blood volumes to be collected during the study are outlined in Table 9.

Table 9 Approximate Total Amount of Blood for Each Subject

| Assessment | Sample Volume<br>(mL) | Number of Samples | Total Blood Volume<br>(mL) |
|---|---|---|---|
| Pharmacokinetics | | | |
| VIS649 | 5 | 16 | 80 |
| Pharmacodynamics | | | |
| Ig | 3.5 | 17 | 59.5 |
| Ig subtypes | 4 | 6 | 24 |
| Lymphocytes (cohorts 1-4) | 14 | 5 | 70 |
| ADA | 5 | 4 | 20 |
| Tetanus/Diphtheria Serology | 7 | 7 | 49 |
| Clinical Laboratory Tests | | | |
| Hematology | 4 | 7 | 28 |
| Clinical chemistry <sup>1</sup> | 8.5 | 4 | 34 |
| Coagulation <sup>2</sup> | 4.5 (+1) | 4 | 22 |
| Total Blood Volume <sup>3</sup> per Subjec | t | | 440.5 |

Abbreviations: ADA: Anti-drug Antibody; Ig: Immunoglobulin; PD: Pharmacodynamics

<sup>&</sup>lt;sup>1</sup> Viral serology and pregnancy tests (women of childbearing potential only) will be performed on the sample collected for clinical chemistry at the Screening Visit.

<sup>&</sup>lt;sup>2</sup> Additional 1mL of blood is collected as a discard tube prior to sample collection.

<sup>&</sup>lt;sup>3</sup> Includes 2 additional follow-up laboratory visits, if needed, per Table 10. Total does exclude repeat and additional laboratory investigations.

### 7. STUDY CONDUCT

#### 7.1. Schedule of Assessments

The study will be comprised of:

- A Screening Visit up to 28 days before dosing
- An in-house stay for approximately 2 to 3 days, with admission to the study center on Day -1, dosing on Day 1 and discharge in the morning of Day 2
- A post-administration period of 16 weeks
- Outpatient visits, on Day 3 (+1 day), 7 (± 1 day), 14, 21, 28, 31 (± 1 day) (cohort 5 only), 35, 42, 49 (cohorts 1-4 only), 56, 70, 84 and 98 (for all visits not otherwise specified, ± 3 days)
- A final Follow-up visit on Day 112 (± 3 days); however, two additional follow-up visits may be performed, at Weeks 20 and 24 post-dosing, if serum immunoglobulins have not returned to > lower limits of normal by the Week 16 (Day 112) visit or if emerging trial data suggest a value of later follow-up (i.e. detection of ADA responses).

The total duration of the clinical study per subject will be up to approximately 20 weeks (5 months), including the Screening period with the possibility of duration extending to 28 weeks (7 months) if follow-ups visits are required. For a detailed Schedule of Assessments, see: Table 10.

Visterra Inc.

Clinical Study Protocol
VIS649-101

CONFIDENTIAL

Table 10 Schedule of Assessments

| Activity | Screen | Base<br>-line | | Post-Dosing Period Assessments | | | | | | | | | | | | litiona<br>'isits <sup>7</sup> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point (Day) | Days - 28<br>to -1 | BL<br>D-1<br>pre-<br>dose | D1 | D2 | D3 | W1/<br>D7 | W2/D<br>14 | W3/D<br>21 | W4/D<br>28 | D31<br>9 | W5/<br>D35 | W6/<br>D42 | W7/<br>D49<br>(coh<br>orts<br>1-4<br>only) | W8/<br>D56 | W10/<br>D70 | W12/<br>D84 | W14/<br>D98 | W16/<br>D112 | W<br>20 | W24 |
| +/- visit allowance | N/A | N/A | N/A | N/A | +1 | +/-1 | +/-3 | +/-3 | +/-3 | +/-1 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/<br>- <b>5</b> | +/-5 |
| In-house Day | | X | X | x <sup>1</sup> | | | | | | | | | | | | | | | | |
| Ambulatory Visit | X | | | | x | X | x | х | X | X | X | X | X | X | X | X | X | X | x <sup>2</sup> | x <sup>2</sup> |
| Procedures | | | | | | | | | | | | | | | | | | | | |
| Informed<br>Consent/HIPAA | х | | | | | | | | | | | | | | | | | | | |
| Verify<br>Inclusion/exclusion<br>criteria | х | х | | | | | | | | | | | | | | | | | | |
| Demographics &<br>Medical History | х | | | | | | | | | | | | | | | | | | | |
| Pregnancy Test<br>(Serum β-hCG) | x | | | | | | | | | | | | | | | | | х | | |
| Pregnancy Test<br>(urine dip stick) | | х | | | | | | | | | | | | | | | | | | |
| Serology -<br>HBsAG, Hepatitis<br>C, HIV-test | х | | | | | | | | | | | | | | | | | | | |
| Drug & alcohol<br>toxicology screen | x | X | | | | | | | | | | | | | | | | | | _ <del>_</del> _ |
| Physical<br>Examination - Full | x | х | | | | | | | | | | | | | | | | | | |
| Physical | | | | | X | | | | x | | | | | X | | x | | x | | <br>I |

Amendment 1, Version 3.0  12 Mar 2019

| Activity | Screen | Base<br>-line | Post-Dosing Period Assessments | | | | | | | | | | | | litiona<br>'isits <sup>7</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point (Day) | Days -<br>28<br>to -1 | BL<br>D-1<br>pre-<br>dose | D1 | D2 | D3 | W1/<br>D7 | W2/D<br>14 | W3/D<br>21 | W4/D<br>28 | D31 | W5/<br>D35 | W6/<br>D42 | W7/<br>D49<br>(coh<br>orts<br>1-4<br>only) | W8/<br>D56 | W10/<br>D70 | W12/<br>D84 | W14/<br>D98 | W16/<br>D112 | W<br>20 | W24 |
| +/- visit allowance | N/A | N/A | N/A | N/A | +1 | +/-1 | +/-3 | +/-3 | +/-3 | +/-1 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/<br>-5 | +/-5 |
| Examination -<br>Brief | | | | | | | | | | | | | | | | | | | | |
| Vital Signs <sup>3</sup> | X | X | X | | X | X | x | | X | | | | | X | | X | | X | | |
| ECG | X | X | x <sup>4</sup> | | | | | | | | | | | | | | | | | |
| Concomitant<br>Medications | X | X | X | | X | X | х | X | X | | X | X | | X | X | X | X | X | X | Х |
| AE Check | | X | X | X | X | X | X | X | X | | X | X | | X | X | X | X | X | X | X |
| IV Study Infusion | | | X | | | | | | | | | | | | | | | | | |
| Laboratory<br>Assessments | | | | | | | | | | | | | | | | | | | | |
| Serum Chemistry /<br>Coagulation | Х | X | | | X | | х | | | | | | | | | | | | | |
| Urinalysis | х | Х | | | х | | | | Х | | | | | Х | | | | Х | | |
| Hematology (CBC with differential) | х | х | | | X | | Х | | х | | | | | х | | х | | | | |
| Blood Sampling<br>for PK <sup>5</sup> | | | <b>x</b> <sup>5</sup> | <b>x</b> <sup>5</sup> | Х | Х | Х | | x <sup>10</sup> | | | Х | | Х | Х | | | Х | | |
| Blood Sampling<br>for PD<br>(Immunoglobulins) | х | X | | | Х | X | х | X | x <sup>10</sup> | | X | X | X | X | X | X | | X | X | X |
| Blood Sampling for Ig subtypes | | Х | | | | Х | | | x <sup>10</sup> | | | | | х | | х | | X | | |
| Blood Sampling | | X | | | | | | | X | | | | | | | | | X | X | X |

Amendment 1, Version 3.0  12 Mar 2019

| Activity | Screen | Base<br>-line | | | | | | J | Post-Dos | ing Pe | riod As | sessmei | nts | | | | | | | litiona<br>'isits <sup>7</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point (Day) | Days -<br>28<br>to -1 | BL<br>D-1<br>pre-<br>dose | D1 | D2 | D3 | W1/<br>D7 | W2/D<br>14 | W3/D<br>21 | W4/D<br>28 | D31 | W5/<br>D35 | W6/<br>D42 | W7/<br>D49<br>(coh<br>orts<br>1-4<br>only) | W8/<br>D56 | W10/<br>D70 | W12/<br>D84 | W14/<br>D98 | W16/<br>D112 | W<br>20 | W24 |
| +/- visit allowance | N/A | N/A | N/A | N/A | +1 | +/-1 | +/-3 | +/-3 | +/-3 | +/-1 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/-3 | +/<br>-5 | +/-5 |
| for PD<br>(lymphocyte<br>populations) <sup>8</sup> | | | | | | | | | | | | | | | | | | | | |
| Blood sampling for | | X | | | | | | | x <sup>10</sup> | | | | | x | | | | x | <b>x</b> <sup>7</sup> | $\mathbf{x}^7$ |
| ADA | | A | | | | | | | | | | | | 1 | | | | A | 71 | |
| Vaccine<br>Administration <sup>9, 10</sup> | | | | | | | | | Х | | | | | | | | | | | |
| Tetanus/diphtheria serology <sup>9, 10</sup> | | | | | | | | | x <sup>10</sup> | Х | X | X | | X | | X | | X | | |

Abbreviations: ADA: Anti-drug Antibody; AE: Adverse event; D: Day; ECG: Electrocardiogram; HBsAG: Hepatitis B surface antigen; HIPAA: Health Insurance Portability and Accountability Act; HIV: Human Immunodeficiency Virus; Ig: Immunoglobulin; IV: Intravenous; N/A: Not Applicable, PD: Pharmacodynamics; PK: Pharmacokinetics; W: Week.

- 1. The first two subjects of each cohort will be discharged 24 hours (Day 2) after the study infusion. All other subjects are discharged on Day 2, 24 hours after study infusion. Discharge from the Phase 1 unit will not occur prior to performing the 24 h post infusion study procedures.
- 2. Optional Visit at Week 20 is only to be made if immunoglobulin levels (IgG, IgM, or IgA) have not returned to normal range by Week 16; the Optional Visit at Week 24 is only to be made if immunoglobulin levels have not returned to normal range by Week 20. If immunoglobulin levels (IgG, IgM, or IgA) have not returned to normal range by Week 16 for one or more subjects, the entire cohort will complete Week 20 and Week 24.
- 3. Vitals signs at Screening and Day -1 will include height and weight, to permit estimated creatinine clearance calculation, as well as blood pressure (bp), heart rate (hr), respiratory rate (rr) and temperature. Subject weight will be measured after admission to the research unit (Day -1) and will be used by

Amendment 1, Version 3.0  12 Mar 2019

pharmacy staff for subject-specific dose calculation. Vital signs at other timepoints will be limited to temperature (Day -1 and Day 1 pre-dose only), bp, hr, and rr. Vital signs measurements on Day 1 will be recorded within 30 minutes prior to the start of the infusion, then every 15 minutes until the infusion is complete and post infusion at 60 minutes, 2 hours and 4 hours. On subsequent visits, vital signs will be recorded, as possible, at approximately the same time of day, if convenient. Post-dose bp should be based on the end of infusion time.

- 4. On Day 1 electrocardiograms will be done within 30 minutes prior to infusion and at the end of the infusion (+10 min).
- 5. On the day of study infusion (Day 1), blood samples for PK analysis will be collected prior to start of the infusion, at the end of infusion (60 minutes), and at 2 hours, 8 hours, and 24 hours post end of infusion. All subjects will have PK samples drawn on Days 3, 7, and Weeks 2 (Day 14), 4 (Day 28), 6 (Day 42), 8 (Day 56), 10 (Day 70), and 16 (112).
- Follow-up visits may be performed if serum immunoglobulin levels or lymphocytes have not returned to > lower limits of normal or if emerging trial data suggest a value of later follow-up (i.e. for ADA responses)
- 9. Activities are only for cohort 5.
- 10. This sampling will be pre-vaccination in cohort 5.

Amendment 1, Version 3.0  12 Mar 2019

#### 7.2. Order of Assessments

The following priority order will be in effect when more than one assessment is required at a pre-dose and post-dose time point, with PK blood sampling being performed nearest to the specified time:

- 1. 12-lead ECG
- 2. Vital signs
- 3. PK blood sampling
- 4. Blood sampling for safety assessments

### 7.3. Early Termination

If a subject withdraws prematurely after dosing, all data normally collected at discharge from the clinical site should be collected at the time of premature discontinuation or at the scheduled discharge. If deemed necessary by the Principal Investigator, the subject will be asked to return at the regularly scheduled End-of-study Visit.

# 7.4. End-of-Study

End-of-study is defined as completion of the final follow-up visit. For those subjects that withdraw prematurely, end-of-study is defined as the time of the subject's last data collection.

#### 7.5. Restrictions

# 7.5.1. Dietary and Fluid Restrictions

**Nicotine** 

Nicotine-containing products (including but not limited to cigarettes, cigars, and chewing or dipping tobacco) is prohibited within less than 3 months before study drug administration. Use of topical or oral nicotine preparations for smoking cessation is also prohibited within less than the past 90 days before study drug administration. Included subjects must abstain from consumption of nicotine-containing products for the duration of the study.

Caffeine:

Consumption of greater than 500 mg of caffeine or xanthine-containing products per day (e.g., coffee, tea, soft drinks, energy drinks, or chocolate) is prohibited. Included subjects must abstain from consuming caffeine or xanthine-containing products from 48 hours prior to check-in on Day -1 through the end of the study.

Alcohol:

Consumption of more than 21 units of alcohol (1 unit of alcohol is equivalent to 8 ounces of beer, 4 ounces of wine, or one ounce of spirits) per week (7 days) is prohibited. Included subjects must abstain from consuming alcohol from 48 hours prior to check-in on Day -1 through the end of the study.

#### 7.5.2. **Other Restrictions**

Medications: Use of prescription or OTC medication is prohibited during the last 30 days or 5 half-lives, whichever is longer, preceding baseline (Day -1) except for acetaminophen, ibuprofen, hormonal contraceptives, topical medications, vitamins, dietary or herbal remedies. Concomitant use of marketed or investigational systemic immunosuppressive or immunomodulatory medications (e.g., corticosteroids, methotrexate, azathioprine, etc. and/or biologics) is prohibited during the last 30 days or 5 half-lives, whichever is longer.

Other:

Blood donation (>500 mL) within 60 days prior to start of Screening and/or donation of any plasma within 7 days prior to baseline (Day-1) and for the duration of the study is prohibited.

# 8. STATISTICAL METHODS

Before database lock, a statistical analysis plan will be issued as a separate document, providing detailed methods for the analyses outlined below. Any deviations from the planned analyses will be described and justified in the CSR.

# **8.1.** Determination of Sample Size

The sample size for this FIH Phase 1 study was not based on formal statistical determinations. The sample size for this study was chosen in consideration of limiting exposure to this new chemical entity while providing sufficient information to evaluate the safety and tolerability of VIS649 in a Phase 1 setting.

# 8.2. Study Population

# 8.2.1. Disposition of Subjects

Subjects entering and completing the clinical study will be listed and summarized using number and percentage.

Subjects excluded from the safety, PK and PD analysis sets and data excluded from the PK and PD analysis sets will be listed including the reason for exclusion. Subject disposition will be summarized. Disposition data will be presented based on all subjects randomized.

#### **8.2.2.** Protocol Deviations

Protocol deviations will be listed by subject.

# 8.2.3. Analysis Populations

- Safety population: All randomized subjects who received at least one dose of study drug. Subjects will be included in the analysis according to the dose and study drug received.
- PK population: All randomized subjects with at least one quantifiable VIS649 concentration. Subjects will be included in the analysis according to the dose and study drug received.
- PD population: The safety population subset with at least one PD parameter assessment (IgA, IgG, IgM) post study drug (VIS649 or placebo) dosing. Subjects will be included in the analysis according to the dose and study drug received.

#### **8.3.** General Considerations

In general, descriptive statistics for continuous variables will be summarized by treatment group using number of subjects, arithmetic mean, standard deviation, median, minimum and maximum; descriptive statistics for categorical data will be summarized by treatment group using frequency counts and percentages. Descriptive statistics for PK parameters will include number of observations, arithmetic mean, standard deviation, arithmetic %CV, and geometric mean, median, geometric %CV, minimum and maximum.

The placebo subjects from cohorts 1-4 will be pooled into a single placebo group for summaries and presentations.

Data grouped by cohorts 1-4, cohort 5 only and overall (all cohorts) will be analyzed separately if deemed appropriate, detail will be described in the SAP.

# 8.4. Demographic and Anthropometric Information and Baseline Characteristics

Demographic and anthropometric variables (age, sex, ethnicity, race, height, weight and BMI) will be listed by subject. Demographic characteristics (age, sex, ethnicity and race) and anthropometric characteristics (height, weight and BMI) will be summarized by treatment and for all subjects in the safety population. The denominator for percentages will be the number of subjects in the safety population for each treatment or for all subjects as applicable.

Medical history data will be listed by subject including visit, description of the disease/procedure, MedDRA System Organ Class (SOC), MedDRA Preferred Term (PT), start date, and stop date (or ongoing if applicable).

#### 8.5. Prior and Concomitant Medication

Prior medications are those that started and stopped prior to the first dose of IMP. Concomitant medications are those taken after first dosing (including medications that started prior to dosing and continued after).

Prior and concomitant medication will be listed by subject and will include the following information: reported name, preferred term, the route of administration, dose, frequency, start date/time, duration and indication.

Prior and concomitant medication will be coded according to the World Health Organization Drug Dictionary latest version.

# 8.6. Drug Administration

A listing of drug administration will be created and will include the date and time of administration. When appropriate, a summary table of compliance will also be created.

# 8.7. Safety Analyses

#### 8.7.1. Adverse Events

Adverse events will be coded using the MedDRA version 21.0 or higher. All AEs will be listed. The incidence of treatment-emergent AEs will be summarized by SOC and PT for each treatment and overall, by severity, and by relationship to IMP.

The categories of the relationship to IMP will be summarized as related (Related, Probably related, and Possibly related) and not related (Unlikely to be related and Unrelated).

Serious AEs will be listed.

Injection site tolerability is defined as AEs demonstrating significant injection site irritation or tissue damage. Injection site tolerability will be reported by treatment group, and time point. The arm used for injection will be listed for subjects in cohort 5.

# 8.7.2. Clinical Laboratory Tests

Individual data listings of laboratory results will be presented for each subject. Flags will be attached to values outside of the laboratory's reference limits along with the Principal Investigator's assessment. Clinically significant laboratory test abnormalities that were considered AEs by the Principal Investigator will be presented in the AE listings.

Clinical laboratory tests (observed values) will be summarized descriptively in tabular format. Safety laboratory data collection should be based on the end of infusion time. Shift tables will be presented for select laboratory parameters.

# 8.7.3. Vital Signs

Individual data listings of vital signs (observed and change from baseline) will be presented for each subject. Individual clinically significant vital signs findings that were considered AEs by the Principal Investigator will be presented in the AE listings.

Observed values as well as change from baseline data will be summarized descriptively in tabular format.

### 8.7.4. Standard 12-lead Electrocardiogram

Standard 12-lead ECG data (observed and change from baseline) will be listed for each subject and time point. Observed values will be classified using frequency counts for normal, abnormality that is not clinically significant, and clinically significant abnormality by dose treatment and time point of collection. Descriptive statistics will be calculated for ECG parameters. The incidence of abnormalities, based on the clinical interpretations from the Principal Investigator, will be enumerated by treatment, and visit. Categorical change from baseline will be summarized descriptively for QTc data.

### 8.7.5. Physical Examination

Abnormal physical examination findings will be listed.

# 8.8. Pharmacokinetics Analyses

VIS649 serum concentrations will be listed by subject.

For cohort 1-4, two sets of summary statistics of VIS649 serum concentrations will be presented by dose level; the first will combine the ethnicities and the second set will stratify each dose level by ethnicity group. Individual and mean VIS649 concentration-time profiles will be plotted for each dose level in both linear and logarithmic scales. Pharmacokinetics parameters will be summarized by dose level for Japanese and non-Japanese subjects using descriptive statistics.



Similar analyses will be applied for data from cohort 5 if deemed appropriate.



# 8.9. Pharmacodynamics Analyses

Pharmacodynamic analysis will be performed using data from all subjects assigned to the PD Population.

PD for circulating lymphocyte, total IgA, IgG and IgM, and other relevant PD applicable markers in serum or appropriate matrix (using the raw data, change from baseline data and % change from baseline, as appropriate) will be summarized and plotted over time. PD should be based on the end of infusion time. Baseline data will be taken as the last measurement prior to dosing or an average of the Screening and baseline values. Further detail will be written in the Statistical Analysis Plan.

#### 8.10. Pharmacokinetics/Pharmacodynamics Analyses



# 8.11. Immunogenicity Data (Antibody to VIS649)

Anti-VIS649 ADA evaluations will be listed including the confirmatory assay (positive/negative). A summary table of the ADA response (positive or negative) will be presented, by treatment (dose of VIS649 or pooled placebo), based on the safety analysis set. In addition, the ADA titers (n, median, minimum and maximum) will be summarized by treatment (dose of VIS649 or pooled placebo) for all subjects with a positive confirmatory assay at each time point; this tabulation will include a summary of the highest titer across all time points for each subject.

#### 8.12. Assessment of Response to Tetanus and Diphtheria Vaccination

Data of assessment of response to tetanus/diphtheria vaccination will be listed by subject for cohort 5.

#### 8.13. Interim Data Reviews

As participants in each dosing cohort complete their Week 16 visit, data clean-up and soft-lock will be performed for cohorts 1-4 only, in order to allow an interim assessment of PK, PD and safety data. PK/PD analysts will be permitted access to unblinded data, to facilitate preparation of blinded data summaries for presentation to the Sponsor. The randomization code will be provided to the bioanalytical laboratories responsible for the analysis PK and PD endpoints. Following analysis of the samples but prior to provision of the data to PAREXEL's statistician, the laboratory will re-code the data back to the corresponding original unique sample ID

numbers, enabling differentiation but not identification of the subjects in order to maintain blinding integrity for the other assessments of the clinical study, until after database lock.

Interim summaries of PK, PD and safety data for entire cohorts (inclusive of both VIS649 and placebo recipients, and therefore, still blinded) may be utilized for various reporting purposes prior to full database lock and unblinding.

# 9. ETHICAL, LEGAL AND ADMINISTRATIVE ASPECTS

# 9.1. Data Quality Assurance

The monitoring of the study will be conducted under the responsibility of the Sponsor by the CRO. The monitor will perform on-site and/or remote monitoring visits as frequently as necessary per the individual study monitoring plan.

The Principal Investigator must prepare and maintain adequate and accurate records of all observations and other data pertinent to the clinical study for each study participant. Frequent communication between the clinical site and the Sponsor is essential to ensure that the safety of the study is monitored adequately. The Principal Investigator will make all appropriate safety assessments on an ongoing basis. The Medical Monitor may review safety information as it becomes available throughout the study.

All aspects of the study will be carefully monitored with respect to Good Clinical Practice (GCP) and SOPs for compliance with applicable government regulations. The Study Monitor will be an authorized individual designated by the Sponsor. The Study Monitor will have access to all records necessary to ensure integrity of the data and will periodically review the progress of the study with the Principal Investigator. The Sponsor will be entitled to audit the facilities used in the clinical and laboratory parts of the study, as well as to access all the data files pertaining to the study. Similar procedures may also be conducted by agents of any regulatory body, either as part of the national GCP compliance program or to review the results of this study in support of a regulatory submission. The Principal Investigator should immediately notify the Sponsor if they have been contacted by a regulatory/ethics agency concerning an inspection.

#### 9.2. Institutional Review Board

Before implementing this study, the protocol, the proposed ICF and HIPAA authorization, and other information given to study volunteers must be reviewed by the IRB of the study site. A signed and dated statement that the protocol and ICF and HIPAA authorization have been approved by the IRB must be given to the Sponsor before study initiation. The name and occupation of the chairperson and the members of the IRB or the IRB's Health and Human Services (assurance number must be supplied to the Sponsor).

#### 9.3. Access to Source Data/Documents

PAREXEL will use an electronic data capture system to manage data collection during this trial. The electronic data capture system (ClinBase) is a software tool designed to ensure quality

assurance and facilitate data capture during clinical trials. Through a system regulated workflow that includes barcode scanning and interfaces to medical equipment to avoid manual data entry, study operations performance is controlled and captured in real time. The system is fully CFR 21 part 11 compliant.

The Principal Investigator will ensure the accuracy, completeness and timeliness of the data reported to the Sponsor. Data collection processes and procedures will be reviewed and validated to ensure completeness, accuracy, reliability and consistency. A complete audit trail will be maintained of all data changes. The Principal Investigator or designee will cooperate with the Sponsor's representative(s) for the periodic review of study documents to ensure the accuracy and completeness of the data capture system at each scheduled monitoring visit.

Electronic consistency checks and manual review will be used to identify any errors or inconsistencies in the data. This information will be provided to the respective study sites by means of electronic or manual queries.

The Principal Investigator or designee will prepare and maintain adequate and accurate study documents (medical records, ECGs, AE and concomitant medication reporting, raw data collection forms, etc.) designed to record all observations and other pertinent data for each subject receiving study drug.

The Principal Investigator will allow Sponsor representatives, contract designees, authorized regulatory authority inspectors and the IRB/IEC to have direct access to all documents pertaining to the study.

# 9.4. Archiving Study Documents

According to ICH SOP guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the study drug. However, these documents should be retained for a longer period if required by the applicable legal requirements.

#### 9.5. Good Clinical Practice

The procedures set out in this clinical study protocol are designed to ensure that the Sponsor and the Principal Investigator abide by the principles of the ICH guidelines on GCP. The clinical study also will be carried out in keeping with national and local legal requirements in accordance with US investigational new drug [IND] regulations [21 CFR 56]).

# 9.6. Informed Consent

Before each subject is enrolled in the clinical study, written informed consent will be obtained from the subject according to the regulatory and legal requirements of the participating country. As part of this procedure, the Principal Investigator must explain orally and in writing the nature, duration and purpose of the study and the action of the drug in such a manner that the subject is aware of the potential risks, inconveniences or AEs that may occur. The subject should be informed that he/she is free to withdraw from the study at any time. He/She will receive all information that is required by federal regulations and ICH guidelines. The Principal Investigator or designee will provide the Sponsor with a copy of the IRB/IEC-approved ICD prior to the start of the study.

The ICD must be signed and dated; one copy will be handed to the subject, and the Principal Investigator will retain a copy as part of the clinical study records. The Principal Investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented.

If a protocol amendment is required, then the ICD may need to be revised to reflect the changes to the protocol. If the ICD is revised, it must be reviewed and approved by the responsible IRB/IEC, and signed by all subjects subsequently enrolled in the clinical study as well as those currently enrolled in the clinical study.

# 9.7. Protocol Approval and Amendment(s)

Before the start of the clinical study, the clinical study protocol and other relevant documents will be approved by the IRB/IEC, in accordance with local legal requirements. The Sponsor must ensure that all ethical and legal requirements have been met before the first subject is enrolled in the clinical study.

This protocol is to be followed exactly. To alter the protocol, amendments must be written, which must be released by the responsible staff and receive IRB/IEC approval prior to implementation (as appropriate).

Administrative changes may be made without the need for a formal amendment, but will also be mentioned in the integrated CSR. All amendments will be distributed to all study protocol recipients, with appropriate instructions.

All protocol deviations will be documented and reported in the final CSR.

# 9.8. Confidentiality Data Protection

All clinical study findings and documents will be regarded as confidential. Study documents (protocols, IBs and other material) will be stored appropriately to ensure their confidentiality. The Principal Investigator and members of his/her research team (including the IRB/IEC) must not disclose such information without prior written approval from the Sponsor, except to the extent necessary to obtain informed consent from subjects who wish to participate in the trial or to comply with regulatory requirements.

The anonymity of participating subjects must be maintained. Subjects will be specified on study documents by their subject number, initial or birth date, not by name. Documents that identify the subject (e.g., the signed ICD) must be maintained in confidence by the Principal Investigator.

# 9.9. Publication Policy

By signing the clinical study protocol, the Principal Investigator agrees with the use of results of the clinical study by the Sponsor for the purposes of national and international registration, publication and information for medical and pharmaceutical professionals. If necessary, the regulatory authorities will be notified of the Principal Investigator's name, address, qualifications and extent of involvement.

The Principal Investigator shall not publish any data (poster, abstract, paper, etc.) without the express written consent of the Sponsor.

#### 10. REFERENCE LIST

- 1. Kiryluk K, Li Y, Scolari F, et al. Discovery of new risk loci for IgA nephropathy implicates genes involved in immunity against intestinal pathogens. *Nat Genet*. 2014; 46(11):1187-1196.
- 2. VIS649 Investigator's Brochure, Version 1.0, dated 15 Aug 2018.
- 3. Yel L. Selective IgA deficiency. J Clin Immunol. 2010; 30(1):10-16.
- 4. Yazdani R, Azizi G, Abolhassani H and Aghamohammadi. Selective IgA deficiency: epidemiology, pathogenesis, clinical phenotype, diagnosis, prognosis and management. *Scand J of Immunol* 2016; 85:3-12.
- 5. Fadlallah J, Kafsi HE, Sterlin D, et al. Microbial ecology perturbation in human IgA deficiency. *Sci. Transl. Med.* 2018; 10(439). pii: eaan1217.
- 6. Furst DE. Serum immunoglobulins and risk of infection: how low can you go? *Semin Arthritis Rheum* 2009; 39(1):18-29.
- 7. Salzer U, Chapel HM, Webster ADB, et al. Mutations in TNFRSF13B encoding TACI are associated with common variable immunodeficiency in humans. *Nat Genet*. 2005; 37:820-828.
- 8. Ameratunga R, Woon ST, Gillis D, Koopmans W, Steele R. New diagnostic criteria for common variable immune deficiency (CVID) which may assist with decisions to treat with intravenous or subcutaneous immunoglobulin. *Clin Exp Immunol* 2013; 174:203-211.
- 9. Ballow M. Primary immunodeficiency disorders: antibody deficiency. *J Allergy Clin Immunol* 2002;109(4):581-591.
- 10. Salzer U, Warnatz K, Peter HH. Common variable immunodeficiency-an update. *Arthritis Research & Therapy* 2012; 14:223-233.
- 11. Full Prescribing Information, Sanofi Pasteur Limited, 420 TENIVAC® (revised April 2013).